CLINICAL TRIAL: NCT01258738
Title: A Multicentre, 12 Week Double Blind Placebo Controlled Randomized Study Of Etanercept On A Background Nsaid In The Treatment Of Adult Subjects With Non Radiographic Axial Spondyloarthritis With A 92 Week Open Label Extension
Brief Title: Study Comparing Etanercept (ETN) Against a Placebo for Etanercept on a Background Nonsteroidal Anti Inflammatory Drug (NSAIDs) in the Treatment of Early Spondyloarthritis (SpA) Patients Who do Not Have X-ray Structural Changes
Acronym: EMBARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1801031; 0881A3-4725 (Other: Alias Study Number); 2010-020077-16 (EudraCT Number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Spondylitis, Ankylosing
Keywords: Early ankylosing spondylitis (SpA) study; efficacy and safety and health out comes
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- etanercept (Active Comparator): In Period 1 : Subjects will receive via a prefilled syringe an active dose equivalent to 1.0ml of Etanercept solution once weekly SC once weekly. Additionally they will continue to take the background non steroidal anti inflammatory drug(NSAID) in the tolerated dose agreed upon by the attending Physician.
  Interventions: Biological: etanercept; Drug: Background NSAID
- PLACEBO (Placebo Comparator): In Period 1: Subjects will receive in a prefilled syringe with a PLACEBO dose equivalent to 1.0 ml of placebo solution once weekly SC Additionally they will continue to take the background non steroidal anti inflammatory drug(NSAID) in the tolerated dose agreed upon by the attending Physician.
  Interventions: Other: PLACEBO; Drug: Background NSAID

INTERVENTIONS:
Biological: etanercept — In Period 1, subjects will receive in a prefilled syringe with 1.0 ml (test article Etanercept (SC) once weekly . Additionally they will continue to take the background non steroidal anti inflammatory drug(NSAID) in the tolerated dose agreed upon by the attending Physician.
  Other Names: ENBREL
  Arms: etanercept
Drug: Background NSAID — Subject will continue to take a concomitant background non steroidal anti inflammatory drug(NSAID)as prescribed by their attending physician. The name and dose of this NSAID is the decision of the attending physician.
  Arms: etanercept
Other: PLACEBO — In Period 1 will receive a prefilled syringe of Placebo for Etanercept Additionally they will continue to take the background non steroidal anti inflammatory drug(NSAID) in the tolerated dose agreed upon by the attending Physician.
  Arms: PLACEBO
Drug: Background NSAID — Subject will continue to take a concomitant background non steroidal anti inflammatory drug(NSAID)as prescribed by attending physician (dose drug selection as tolerated and agreed upon by the attending Physician).
  Arms: PLACEBO

SUMMARY:
This is a two part study. During period one there will be a comparison of Etanercept (ETN) against a placebo with both arms maintaining the background anti inflammatory drug prescribed by their Physician. The hypothesis is that Etanercept will be superior to the placebo arm as determined by the proportion of subjects achieving Assessments in Ankylosing Spondylitis (ASAS)40 improvement at 12 weeks. This will be followed by 92 weeks extension where everyone in the trial receives Etanercept (ETN) and a background non steroidal anti inflammatory drug(NSAID).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of axial spondyloarthritis as defined by Assessments in Ankylosing Spondylitis (ASAS)criteria
* Active symptoms defined as Ankylosing Spondylitis Disease Activity Index{BASDAI) > or = 4
* Axial symptoms of back pain with a less than favorable response to on steroidal anti inflammatory drugs at optimal dosage for greater than 4 weeks

Exclusion Criteria:

* Evidence of current or recent episode of uveitis
* Evidence of IBD flare within 6 months
* Previous treatment with an anti Tumor necrosis factor(TNF)
* Active tuberculosis
* Radiographic sacroiliitis grade 3-4 unilaterally or >= 2 bilaterally

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- Argentina (2):
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Consultorios Reumatológicos Pampa, Buenos Aires
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent
  - Reuma Instituut, Hasselt
  - AZ Groeninge, Kortrijk
- Colombia (3):
  - Preventive Care Ltda., Chía, Cundinamarca
  - Ips Medicity S.A.S, Bucaramanga, Santander Department
  - Servimed Sas, Bucaramanga, Santander Department
- Czechia (3):
  - Revmatologicky ustav, Prague
  - Mediscan Group, s.r.o., Praha 11 - Chodov
  - Medical Plus s.r.o., Uherské Hradiště
- Finland (2):
  - Meilahden kolmiosairaala, Helsinki
  - Kiljavan Lääketutkimus, Hyvinkää
- France (4):
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - CHU Lapeyronie, Immuno-Rhumatologie, Montpellier
  - Hôpital Cochin, Paris
  - CHU de Tours, Tours
- Germany (5):
  - Charite - Campus Benjamin Franklin, Medizinische Klinik I - Rheumatologie, Berlin
  - Studienambulanz, Medizinische Klinik 3, Universitaetsklinikum Erlangen, Erlangen
  - Schoen Klinik Hamburg-Eilbek, Abt. Rheumatologie und Klin. Immunologie, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - MEDIGREIF Verwaltungs- und Betriebsgesellschaft Fachkrankenhaus Vogelsang-Gommern mbH, Vogelsang-Gommern
- Hungary (6):
  - Budai Irgalmasrendi Korhaz, Budapest, Budapest
  - Orszagos Reumatologiai es Fizioterapias Intezet/Klinikai Immunologiai es Reumatologiai Osztaly, Budapest
  - Qualiclinic Egeszsegugyi Szolgaltato es Kutatasszervezo Kft., Budapest
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft., Budapest
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
  - Csolnoky Ferenc Korhaz, Veszprém
- Netherlands (2):
  - Academic Medical Centre (AMC) / Division of Clinical Immunology and Rheumatology, Amsterdam, North Holland
  - Leiden University Medical Center, Reumatologie, Leiden
- Russia (5):
  - Rheumatology Research Institute of Russian Academy of Medical Sciences, Moscow
  - Russian Cardiology Research-and-Production Complex, Moscow
  - Saint-Petersburg State Budgetary Healthcare Institution, Saint Petersburg
  - Limited Liability Company NMC Tomography, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
- South Korea (3):
  - Gachon University Gil Hospital, Incheon, Gwangyeogsiv
  - Chonnam National University Hospital, Gwangju
  - Hanyang University Hospital, Seoul
- Spain (4):
  - Hospital Virgen Macarena, Seville, Andalusia
  - Hospital Reina Sofia, Córdoba, Cordoba
  - Complexo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid
- Taiwan (3):
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Rhuematology Clinical Research Unit, Cambridge, Cambridgeshire
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hants.
  - Norfolk and Norwich University Hospital NHS Trust, Norwich, Norfolk
  - Russells Hall Hospital, Dudley, West Midlands
  - Whipps Cross University Hospital,, London

REFERENCES:
- [Derived] Maksymowych WP, Claudepierre P, de Hooge M, Lambert RG, Landewe R, Molto A, van der Heijde D, Bukowski JF, Jones H, Pedersen R, Szumski A, Vlahos B, Dougados M. Erosions on T1-Weighted Magnetic Resonance Imaging Versus Radiography of Sacroiliac Joints in Recent-Onset Axial Spondyloarthritis: 2-Year Data (EMBARK Trial and DESIR Cohort). J Rheumatol. 2024 May 1;51(5):462-471. doi: 10.3899/jrheum.2023-0906. PMID 38359938
- [Derived] Schneeberger EE, Citera G, de Leon DP, Szumski AE, Kwok K, Cutri M, Dougados M. Simplified Ankylosing Spondylitis Disease Activity Score (SASDAS) Versus ASDAS: A Post Hoc Analysis of a Randomized Controlled Trial. J Rheumatol. 2022 Oct;49(10):1100-1108. doi: 10.3899/jrheum.211075. Epub 2022 Jul 15. PMID 35840157
- [Derived] Maksymowych WP, Claudepierre P, de Hooge M, Lambert RG, Landewe R, Molto A, van der Heijde D, Bukowski JF, Jones H, Pedersen R, Szumski A, Vlahos B, Dougados M. Structural changes in the sacroiliac joint on MRI and relationship to ASDAS inactive disease in axial spondyloarthritis: a 2-year study comparing treatment with etanercept in EMBARK to a contemporary control cohort in DESIR. Arthritis Res Ther. 2021 Jan 29;23(1):43. doi: 10.1186/s13075-021-02428-8. PMID 33514428
- [Derived] Dougados M, van der Heijde D, Tsai WC, Saaibi D, Marshall L, Jones H, Pedersen R, Vlahos B, Tarallo M. Relationship between disease activity status or clinical response and patient-reported outcomes in patients with non-radiographic axial spondyloarthritis: 104-week results from the randomized controlled EMBARK study. Health Qual Life Outcomes. 2020 Jan 3;18(1):4. doi: 10.1186/s12955-019-1260-4. PMID 31900174
- [Derived] Dougados M, Maksymowych WP, Landewe RBM, Molto A, Claudepierre P, de Hooge M, Lambert RG, Bonin R, Bukowski JF, Jones HE, Logeart I, Pedersen R, Szumski A, Vlahos B, van der Heijde D. Evaluation of the change in structural radiographic sacroiliac joint damage after 2 years of etanercept therapy (EMBARK trial) in comparison to a contemporary control cohort (DESIR cohort) in recent onset axial spondyloarthritis. Ann Rheum Dis. 2018 Feb;77(2):221-227. doi: 10.1136/annrheumdis-2017-212008. Epub 2017 Sep 29. PMID 28970213
- [Derived] Maksymowych WP, Wichuk S, Dougados M, Jones HE, Pedersen R, Szumski A, Marshall L, Bukowski JF, Lambert RG. Modification of structural lesions on MRI of the sacroiliac joints by etanercept in the EMBARK trial: a 12-week randomised placebo-controlled trial in patients with non-radiographic axial spondyloarthritis. Ann Rheum Dis. 2018 Jan;77(1):78-84. doi: 10.1136/annrheumdis-2017-211605. Epub 2017 Sep 29. PMID 28970212
- [Derived] Brown MA, Bird PA, Robinson PC, Mease PJ, Bosch FVD, Surian C, Jones H, Szumski A, Marshall L, Wiid Z, Dougados M. Evaluation of the effect of baseline MRI sacroiliitis and C reactive protein status on etanercept treatment response in non-radiographic axial spondyloarthritis: a post hoc analysis of the EMBARK study. Ann Rheum Dis. 2018 Jul;77(7):1091-1093. doi: 10.1136/annrheumdis-2017-211313. Epub 2017 Jul 3. No abstract available. PMID 28673924
- [Derived] Maksymowych WP, Wichuk S, Dougados M, Jones H, Szumski A, Bukowski JF, Marshall L, Lambert RG. MRI evidence of structural changes in the sacroiliac joints of patients with non-radiographic axial spondyloarthritis even in the absence of MRI inflammation. Arthritis Res Ther. 2017 Jun 6;19(1):126. doi: 10.1186/s13075-017-1342-9. PMID 28587658
- [Derived] Dougados M, van der Heijde D, Sieper J, Braun J, Citera G, Lenaerts J, van den Bosch F, Wei JC, Pedersen R, Bonin R, Jones H, Marshall L, Logeart I, Vlahos B, Bukowski JF, Maksymowych WP. Effects of Long-Term Etanercept Treatment on Clinical Outcomes and Objective Signs of Inflammation in Early Nonradiographic Axial Spondyloarthritis: 104-Week Results From a Randomized, Placebo-Controlled Study. Arthritis Care Res (Hoboken). 2017 Oct;69(10):1590-1598. doi: 10.1002/acr.23276. Epub 2017 Aug 31. PMID 28482137
- [Derived] Maksymowych WP, Dougados M, van der Heijde D, Sieper J, Braun J, Citera G, Van den Bosch F, Logeart I, Wajdula J, Jones H, Marshall L, Bonin R, Pedersen R, Vlahos B, Kotak S, Bukowski JF. Clinical and MRI responses to etanercept in early non-radiographic axial spondyloarthritis: 48-week results from the EMBARK study. Ann Rheum Dis. 2016 Jul;75(7):1328-35. doi: 10.1136/annrheumdis-2015-207596. Epub 2015 Aug 12. PMID 26269397
- [Derived] Dougados M, van der Heijde D, Sieper J, Braun J, Maksymowych WP, Citera G, Miceli-Richard C, Wei JC, Pedersen R, Bonin R, Rahman MU, Logeart I, Wajdula J, Koenig AS, Vlahos B, Alvarez D, Bukowski JF. Symptomatic efficacy of etanercept and its effects on objective signs of inflammation in early nonradiographic axial spondyloarthritis: a multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Rheumatol. 2014 Aug;66(8):2091-102. doi: 10.1002/art.38721. PMID 24891317
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801031&StudyName=Study%20Comparing%20Etanercept%20%28ETN%29%20Against%20a%20Placebo%20for%20Etanercept%20on%20a%20Background%20Nonsteroidal%20Anti%20Inflammatory%20Drug%20%28NSAIDs%29%20in%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 48 centers in 14 countries.
Pre-assignment Details: Eligible participants were randomized to receive etanercept or placebo for 12 week controlled (double-blind) period. Participants completing 12 week period entered a 92 week open-label period.
Groups:
- Etanercept: Participants were treated with etanercept subcutaneous injection weekly plus stable background non-steroidal anti-inflammatory drug (NSAID) at optimal anti-inflammatory dose for 12 weeks (double-blind period). All participants who completed the 12-week double-blind period entered into a 92 week open-label period and received etanercept 50 mg once weekly and background NSAID.
- Placebo: Participants were treated with placebo subcutaneous injection weekly plus stable background NSAID at optimal anti-inflammatory dose for 12 weeks (double-blind period). All participants who completed the 12-week double-blind period entered into a 92 week open-label period and received etanercept 50 mg once weekly and background NSAID.
Period: Double-blind Period
Arm/Group | Etanercept | Placebo
Started | 111 | 114
Treated | 111 | 113
Completed | 102 | 107 (Only 106 participants entered the open label period.)
Not Completed | 9 | 7
Not completed — Did not meet inclusion criteria | 3 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Adverse Event | 3 | 1
Period: Open-label Period
Arm/Group | Etanercept | Placebo
Started | 102 | 106
Completed | 85 | 85
Not Completed | 17 | 21
Not completed — Did not meet inclusion criteria | 0 | 1
Not completed — Insufficient clinical response | 5 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 4 | 5
Not completed — Other Reasons | 0 | 1
Not completed — Withdrawn due to pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set for the double blind period was defined as all randomized participants who took at least one dose of study medication. A total of 224 of the 225 randomized participants received study medication (1 subject randomized to the placebo group did not receive study medication).
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 111 | 113 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (7.8) | 32.0 (7.8) | 31.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 50 | 91
  Male | 70 | 63 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Ankylosing Spondylitis (ASAS) 40 Response at Week 12
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) in 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement from baseline and an absolute change ≥ 20 units on a 0-100 scale (0 = no disease activity, 100 = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Week 12
Population: Modified intent-to-treat (mITT) population defined as all randomized participants who took at least one dose of study drug, had at least one on-therapy evaluation and met the ASAS classification criteria for axial spondyloarthritis (AxSpA). Missing data were imputed through last observation carried forward (LOCF) approach.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
Percentage of participants | 32.38 | 15.74
Statistical Analysis 1: Comparison: Etanercept vs Placebo; The null hypothesis was that the efficacy of etanercept was not different from placebo as measured by the proportion of subjects achieving an ASAS 40 response after 12 weeks of treatment. The alternative hypothesis was that the efficacy of etanercept was different from placebo. The primary endpoint was tested at 2-sided alpha = 0.05 significance level. Comparative analysis was carried out for Week 12 data only; Test type: Superiority or Other; p = 0.0062, Cochran-Mantel-Haenszel — P-value <0.05 was required to declare statistical significance; Mean Difference (Final Values) = 16.64, 95% CI 2-sided [5.36 to 27.92]

2. Secondary Outcome: Percentage of Participants Achieving ASAS 40 Response at Time Points
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 40 = 40% improvement from baseline and an absolute change ≥ 20 units on a 0-100 scale (0 = no disease activity, 100 = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Baseline to Week 104
Population: mITT population defined as all randomized participants who took at least one dose of study drug, had at least one on-therapy evaluation and met the ASAS classification criteria for AxSpA. Missing data were imputed through LOCF approach.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
Percentage of participants
  Week 2 (N=105, 106) | 15.24 | 3.77
  Week 4 (N=105, 108) | 20.00 | 14.81
  Week 8 (N=105, 108) | 28.57 | 15.74
  Week 12 (N= 105, 108) | 33.33 | 14.81
  Week 16 (N= 100, 105) | 42.00 | 38.10
  Week 24 (N= 100, 105) | 44.00 | 51.43
  Week 32 (N= 100, 105) | 47.00 | 52.38
  Week 40 (N= 100, 105) | 55.00 | 53.33
  Week 48 (N= 100, 105) | 52.00 | 53.33
  Week 56 (N= 100, 105) | 52.00 | 59.05
  Week 68 (N= 100, 105) | 54.00 | 58.10
  Week 80 (N= 100, 105) | 49.00 | 58.10
  Week 92 (N= 100, 105) | 57.00 | 61.90
  Week 104 (N= 100, 105) | 56.00 | 61.90
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 2; Test type: Superiority or Other; p = 0.0059, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 11.46, 95% CI 2-sided [3.69 to 19.24]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 4; Test type: Superiority or Other; p = 0.3786, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 5.19, 95% CI 2-sided [-4.98 to 15.35]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 8; Test type: Superiority or Other; p = 0.0304, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.83, 95% CI 2-sided [1.79 to 23.87]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 12; Test type: Superiority or Other; p = 0.0023, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.52, 95% CI 2-sided [7.29 to 29.75]

3. Secondary Outcome: Percentage of Participants Achieving ASAS 20 Response at Time Points
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement from baseline and an absolute change ≥ 10 units on a 0-100 scale (0=no disease activity; 100 = high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
Percentage of participants
  Week 2 (N = 105, 106) | 30.48 | 16.04
  Week 4 (N = 105, 108) | 37.14 | 26.85
  Week 8 (N = 105, 108) | 48.57 | 37.96
  Week 12 (N = 105, 109) | 52.38 | 36.70
  Week 16 (N= 100, 105) | 64.00 | 65.71
  Week 24 (N = 100, 105) | 65.00 | 71.43
  Week 32 (N = 100, 105) | 64.00 | 71.43
  Week 40 (N = 100, 105) | 73.00 | 73.33
  Week 48 (N = 100, 105) | 71.00 | 72.38
  Week 56 (N = 100, 105) | 70.00 | 76.19
  Week 68 (N = 100, 105) | 69.00 | 76.19
  Week 80 (N = 100, 105) | 65.00 | 70.48
  Week 92 (N = 100, 105) | 71.00 | 74.29
  Week 104 (N = 100, 105) | 70.00 | 79.05
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0189, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.44, 95% CI 2-sided [3.20 to 25.68]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0983, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.29, 95% CI 2-sided [-2.17 to 22.75]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0867, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 10.61, 95% CI 2-sided [-2.63 to 23.84]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0195, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 16.27, 95% CI 2-sided [3.10 to 29.43]

4. Secondary Outcome: Percentage of Participants Achieving ASAS 5/6 Response at Time Points
Description: ASAS 5/6 consists of 6 domains: the 4 used in ASAS 20 (participant global assessment of disease activity, pain, function, inflammation measured on a 0-100 scale, where 0 = no disease activity and 100 = high disease activity) plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). Achieving ASAS 5/6 requires a 20% improvement compared to baseline in ≥ 5 domains and no worsening in the remaining domain.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
Percentage of participants
  Week 2 (N = 102, 105) | 15.69 | 2.86
  Week 4 (N = 103, 107) | 23.30 | 8.41
  Week 8 (N = 103, 107) | 33.01 | 11.21
  Week 12 (N = 105, 109) | 33.01 | 10.38
  Week 16 (N = 100, 105) | 37.00 | 34.29
  Week 24 (N = 100, 105) | 41.00 | 42.86
  Week 32 (N = 100, 105) | 40.00 | 40.95
  Week 40 (N = 100, 105) | 45.00 | 40.95
  Week 48 (N = 100, 105) | 49.00 | 45.71
  Week 56 (N = 100, 105) | 42.00 | 45.71
  Week 68 (N = 100, 105) | 42.00 | 43.81
  Week 80 (N = 100, 105) | 39.00 | 37.14
  Week 92 (N = 100, 105) | 46.00 | 47.62
  Week 104 (N = 100, 105) | 43.00 | 40.95
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 22.63, 95% CI 2-sided [11.85 to 33.41]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0021, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.83, 95% CI 2-sided [5.09 to 20.57]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0020, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 14.89, 95% CI 2-sided [5.18 to 24.60]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 21.79, 95% CI 2-sided [10.92 to 32.67]

5. Secondary Outcome: Mean Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) High Sensitivity CRP (hsCRP) Score at Time Points
Description: ASDAS includes CRP (mg/L) or ESR (mm/hr); Apart from the value of CRP or ESR, the four additional self-reported items (rated on 0-10cm VAS or 0-10 numerical rating scale [NRS]) included in this index are back pain, duration of morning stiffness, peripheral pain/swelling and patient global assessment of disease activity. The ASDAS scores are then calculated as follows: ASDAS_CRP = (0.121 x total back pain) + (0.110 x subject global) + (0.073 x peripheral pain/swelling) + (0.058 x duration of morning stiffness) + (0.579 x Ln(CRP+1)). And ASDAS_ESR: (0.079 x total back pain) + (0.113 x subject global) + (0.086 x peripheral pain/swelling) + (0.069 x duration of morning stiffness) + (0.293 x √ESR). In addition, the proportion of participants who achieve inactive disease based on the ASDAS will be determined for each group. Inactive disease is defined as an ASDAS score <1.3.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
Units on a scale
  Week 2 (N = 104, 106) | -0.74 (0.10) | -0.20 (0.10)
  Week 4 (N = 104, 108) | -0.92 (0.11) | -0.30 (0.10)
  Week 8 (N = 104, 108) | -1.09 (0.13) | -0.48 (0.12)
  Week 12 (N= 104, 108) | -1.27 (0.11) | -0.63 (0.08)
  Week 16 (N= 99, 104) | -1.41 (0.11) | -1.35 (0.11)
  Week 24 (N= 99, 104) | -1.48 (0.11) | -1.55 (0.11)
  Week 32 (N= 99, 104) | -1.44 (0.11) | -1.52 (0.11)
  Week 40 (N= 99, 104) | -1.64 (0.11) | -1.60 (0.12)
  Week 48 (N= 99, 104) | -1.62 (0.11) | -1.63 (0.12)
  Week 56 (N= 99, 104) | -1.61 (0.12) | -1.65 (0.11)
  Week 68 (N= 99, 104) | -1.60 (0.11) | -1.65 (0.11)
  Week 80 (N= 99, 104) | -1.53 (0.12) | -1.61 (0.12)
  Week 92 (N= 99, 104) | -1.63 (0.12) | -1.70 (0.12)
  Week 104 (N= 99, 104) | -1.59 (0.12) | -1.68 (0.12)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test. For open-label period results include unadjusted mean changes and standard errors, no covariate adjustments were applied; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.74 to -0.34]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.81 to -0.41]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.85 to -0.37]

6. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission at Time Points
Description: Partial remission defined as a score of 20 units or less (on a scale of 0-100, where 0 = no disease activity and 100 = high disease activity) in each of the 4 Assessment in ASAS domains: participant global assessment of disease activity, pain, function, and inflammation. For scale, 100 = high disease activity.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
Percentage of participants
  Week 2 (N = 105, 108) | 11.43 | 2.78
  Week 4 (N = 105, 109) | 10.48 | 3.67
  Week 8 (N = 105, 109) | 21.90 | 9.17
  Week 12 (N = 105, 109) | 24.76 | 11.93
  Week 16 (N = 100, 105) | 29.00 | 28.57
  Week 24 (N = 100, 105) | 32.00 | 42.86
  Week 32 (N = 100, 105) | 28.00 | 41.90
  Week 40 (N = 100, 105) | 40.00 | 45.71
  Week 48 (N = 100, 105) | 38.00 | 37.14
  Week 56 (N = 100, 105) | 40.00 | 43.81
  Week 68 (N = 100, 105) | 37.00 | 48.57
  Week 80 (N = 100, 105) | 34.00 | 49.52
  Week 92 (N = 100, 105) | 39.00 | 49.52
  Week 104 (N = 100, 105) | 40.00 | 57.14
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0209, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.84, 95% CI 2-sided [2.58 to 23.09]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0179, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.65, 95% CI 2-sided [1.82 to 15.48]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0611, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 6.81, 95% CI 2-sided [-0.03 to 13.65]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0141, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 12.73, 95% CI 2-sided [3.14 to 22.32]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Time to ASAS Partial Remission
Description: The median time to partial remission was not reached at Week 12. Hence, we report an estimate of the percentage of participants, estimated using Kaplan-Meier approach.
Time Frame: Week 12
Population: mITT population defined as all randomized participants who took at least one dose of study drug, had at least one on-therapy evaluation and met the ASAS classification criteria for AxSpA.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
percentage of participants | 43.3 [30.4 to 59.0] | 22.3 [12.5 to 38.1]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 12 data only; Test type: Superiority or Other; p = 0.0022, Log Rank

8. Secondary Outcome: Mean Change From Baseline in Visual Analogue Scale (VAS) Physician Global Assessments at Time Points
Description: The Investigator estimated the participant's overall disease activity over the previous 48 hours (this was independent of the Subject Assessment of Disease Activity) using a scale between 0 mm (none) and 100 mm (severe).
Time Frame: Baseline to Week 104
Population: mITT population defined as all randomized participants who took at least one dose of study drug, had at least one on-therapy evaluation and met the ASAS classification criteria for AxSpA. Missing data were imputed through LOCF approach. The values were converted to cm for analysis purposes.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 102 | 105
cm
  Week 2 (N = 101, 104) | -1.40 (0.24) | -0.80 (0.23)
  Week 4 (N = 101, 105) | -1.91 (0.25) | -1.49 (0.24)
  Week 8 (N = 101, 105) | -2.39 (0.27) | -2.10 (0.25)
  Week 12 (N = 100, 105) | -2.74 (0.29) | -2.04 (0.28)
  Week 16 (N = 96, 101) | -3.36 (0.23) | -2.78 (0.23)
  Week 24 (N = 96, 101) | -3.66 (0.20) | -3.25 (0.23)
  Week 32 (N = 96, 101) | -3.66 (0.21) | -3.38 (0.22)
  Week 40 (N = 96, 101) | -3.83 (0.21) | -3.44 (0.21)
  Week 48 (N = 96, 101) | -3.93 (0.23) | -3.53 (0.21)
  Week 56 (N = 96, 101) | -3.98 (0.24) | -3.67 (0.22)
  Week 68 (N = 96, 101) | -3.98 (0.22) | -3.60 (0.22)
  Week 80 (N = 96, 101) | -4.03 (0.22) | -3.54 (0.24)
  Week 92 (N = 96, 101) | -4.00 (0.22) | -3.43 (0.24)
  Week 104 (N = 96, 101) | -4.12 (0.23) | -3.78 (0.22)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0156, ANCOVA; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.26 to -0.13]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0111, ANCOVA; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.06 to -0.14]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0936, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.91 to 0.07]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.2678, ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.81 to 0.23]

9. Secondary Outcome: Mean Change From Baseline in VAS Score for Subject Assessment of Disease Activity at Time Points
Description: Participants to assess their overall disease activity over the last 48 hours using a pain scale between 0 mm (none) and 100 mm (severe), which corresponded to the magnitude of their pain.
Time Frame: Baseline to Week 104
Population: as for outcome 8
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
cm
  Week 2 (N = 105, 108) | -1.00 (0.27) | -0.08 (0.26)
  Week 4 (N = 105, 109) | -1.34 (0.29) | -0.55 (0.27)
  Week 8 (N = 105, 109) | -1.85 (0.32) | -1.02 (0.30)
  Week 12 (N = 105, 109) | -2.06 (0.31) | -1.26 (0.30)
  Week 16 (N = 100, 105) | -2.81 (0.27) | -2.65 (0.24)
  Week 24 (N = 100, 105) | -2.92 (0.28) | -3.21 (0.23)
  Week 32 (N = 100, 105) | -2.99 (0.27) | -3.23 (0.27)
  Week 40 (N = 100, 105) | -3.38 (0.27) | -3.33 (0.25)
  Week 48 (N = 100, 105) | -3.24 (0.28) | -3.36 (0.27)
  Week 56 (N = 100, 105) | -3.30 (0.28) | -3.45 (0.25)
  Week 68 (N = 100, 105) | -3.31 (0.28) | -3.57 (0.25)
  Week 80 (N = 100, 105) | -3.10 (0.27) | -3.49 (0.25)
  Week 92 (N = 100, 105) | -3.34 (0.28) | -3.65 (0.25)
  Week 104 (N = 100, 105) | -3.33 (0.30) | -3.75 (0.24)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test. For open-label period results included unadjusted mean changes and standard errors, no covariate adjustments were applied; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0102, ANCOVA; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.40 to -0.19]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.44 to -0.39]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0057, ANCOVA; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.35 to -0.23]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0077, ANCOVA; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.44 to -0.22]

10. Secondary Outcome: Changes From Baseline in VAS Score for Nocturnal Back Pain at Time Points
Description: The VAS scale was used to assess the level of nocturnal pain during the past 48 hours. For this, participants marked their level of pain on a 100 mm VAS anchored by 0 for "No pain " to 100 mm for "Most Severe Pain."
Time Frame: Baseline to Week 104
Population: as for outcome 8
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
cm
  Week 2 (N = 105, 107) | -1.10 (0.31) | -0.31 (0.29)
  Week 4 (N = 105, 109) | -1.54 (0.33) | -0.71 (0.31)
  Week 8 (N = 105, 109) | -2.31 (0.33) | -1.34 (0.31)
  Week 12 (N = 105, 109) | -1.96 (0.36) | -1.03 (0.34)
  Week 16 (N = 100, 105) | -2.97 (0.31) | -2.63 (0.26)
  Week 24 (N = 100, 105) | -2.79 (0.30) | -3.25 (0.26)
  Week 32 (N = 100, 105) | -2.69 (0.31) | -3.11 (0.29)
  Week 40 (N = 100, 105) | -3.34 (0.31) | -3.30 (0.26)
  Week 48 (N = 100, 105) | -3.22 (0.31) | -3.21 (0.27)
  Week 56 (N = 100, 105) | -3.15 (0.33) | -3.40 (0.27)
  Week 68 (N = 100, 105) | -3.07 (0.33) | -3.27 (0.26)
  Week 80 (N = 100, 105) | -3.01 (0.31) | -3.32 (0.27)
  Week 92 (N = 100, 105) | -3.26 (0.32) | -3.43 (0.27)
  Week 104 (N = 100, 105) | -3.28 (0.34) | -3.59 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0091, ANCOVA; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.62 to -0.23]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0097, ANCOVA; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.38 to -0.19]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0101, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.45 to -0.20]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0031, ANCOVA; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.61 to -0.33]

11. Secondary Outcome: Changes From Baseline in VAS Score for Total Back Pain at Time Points
Description: The VAS scale was used to assess the level of total back pain during the past 48 hours. For this, participants marked their level of pain on a 100 mm VAS anchored by 0 for "No pain " to 100 mm for "Most Severe Pain."
Time Frame: Baseline to Week 104
Population: as for outcome 8
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
cm
  Week 2 (N = 105, 107) | -0.95 (0.29) | -0.37 (0.27)
  Week 4 (N = 105, 109) | -1.52 (0.31) | -0.88 (0.29)
  Week 8 (N = 105, 109) | -2.19 (0.33) | -1.18 (0.31)
  Week 12 (n = 105, 109) | -2.32 (0.28) | -1.39 (0.21)
  Week 16 (n = 100, 105) | -2.73 (0.29) | -2.64 (0.25)
  Week 24 (n = 100, 105) | -2.76 (0.28) | -2.92 (0.24)
  Week 32 (n = 100, 105) | -2.58 (0.29) | -2.87 (0.26)
  Week 40 (n = 100, 105) | -3.30 (0.28) | -3.20 (0.24)
  Week 48 (n = 100, 105) | -3.09 (0.29) | -3.14 (0.25)
  Week 56 (n = 100, 105) | -3.10 (0.29) | -3.17 (0.26)
  Week 68 (n = 100, 105) | -3.02 (0.31) | -3.23 (0.26)
  Week 80 (n = 100, 105) | -2.95 (0.29) | -3.17 (0.26)
  Week 92 (n = 100, 105) | -3.30 (0.29) | -3.33 (0.27)
  Week 104 (n = 100, 105) | -3.22 (0.32) | -3.47 (0.26)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0064, ANCOVA; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.49 to -0.25]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0407, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.12 to -0.02]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0349, ANCOVA; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.24 to -0.05]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0021, ANCOVA; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-1.65 to -0.37]

12. Secondary Outcome: Changes From Baseline in the Bath Ankylosing Spondylitis Functional Index (BASFI) Total Score at Time Points
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in AS. Utilizing a VAS of 0-10 (0 = easy, 10 = impossible), participants answered 10 questions assessing their ability in completing normal daily activities or physically demanding activities. The BASFI score is a mean score of the 10 questions.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N = 105, 107) | -0.82 (0.21) | -0.27 (0.20)
  Week 4 (N = 105, 108) | -0.99 (0.22) | -0.44 (0.21)
  Week 8 (N = 105, 108) | -1.28 (0.23) | -0.73 (0.22)
  Week 12 (N = 105, 109) | -1.41 (0.24) | -0.84 (0.23)
  Week 16 (N = 100, 105) | -1.78 (0.23) | -1.75 (0.19)
  Week 24 (N = 100, 105) | -1.89 (0.22) | -1.85 (0.20)
  Week 32 (N = 100, 105) | -1.81 (0.22) | -1.98 (0.21)
  Week 40 (N = 100, 105) | -2.19 (0.23) | -2.13 (0.21)
  Week 48 (N = 100, 105) | -2.19 (0.23) | -2.10 (0.22)
  Week 56 (N = 100, 105) | -2.15 (0.22) | -2.30 (0.21)
  Week 68 (N = 100, 105) | -2.21 (0.21) | -2.31 (0.22)
  Week 80 (N = 100, 105) | -2.23 (0.21) | -2.19 (0.22)
  Week 92 (N = 100, 105) | -2.31 (0.23) | -2.35 (0.22)
  Week 104 (N = 100, 105) | -2.40 (0.23) | -2.36 (0.23)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0164, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.04 to -0.11]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0095, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.95 to -0.13]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0127, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.99 to -0.12]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0166, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.99 to -0.10]

13. Secondary Outcome: Mean Change From Baseline in BASFI Full Day Activities at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 104, 107) | -0.99 (0.26) | -0.21 (0.25)
  Week 4 (N= 104, 108) | -1.37 (0.28) | -0.70 (0.26)
  Week 8 (N= 104, 108) | -1.80 (0.27) | -1.05 (0.26)
  Week 12 (N = 104, 108) | -2.11 (0.29) | -1.16 (0.27)
  Week 16 (N = 99, 105) | -2.37 (0.25) | -2.03 (0.24)
  Week 24 (N = 99, 105) | -2.42 (0.25) | -2.13 (0.25)
  Week 32 (N = 99, 105) | -2.43 (0.23) | -2.38 (0.25)
  Week 40 (N = 99, 105) | -2.93 (0.26) | -2.30 (0.25)
  Week 48 (N = 99, 105) | -2.73 (0.25) | -2.34 (0.27)
  Week 56 (N = 99, 105) | -2.66 (0.25) | -2.59 (0.26)
  Week 68 (N = 99, 105) | -2.82 (0.25) | -2.71 (0.27)
  Week 80 (N = 99, 105) | -2.75 (0.25) | -2.58 (0.27)
  Week 92 (N = 99, 105) | -2.93 (0.27) | -2.70 (0.27)
  Week 104 (N = 99, 105) | -3.04 (0.27) | -2.66 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0029, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.28 to -0.27]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0147, ANCOVA; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.21 to -0.13]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0056, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.28 to -0.22]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0010, ANCOVA; Mean Difference (Final Values) = -0.95, 95% CI 2-sided [-1.52 to -0.39]

14. Secondary Outcome: Mean Change From Baseline in BASFI Bending Forward at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -1.05 (0.28) | -0.40 (0.26)
  Week 4 (N= 105, 108) | -0.96 (0.29) | -0.56 (0.28)
  Week 8 (N= 105, 108) | -1.34 (0.29) | -0.65 (0.27)
  Week 12 (N = 105, 109) | -1.34 (0.29) | -0.85 (0.27)
  Week 16 (N = 100, 105) | -1.76 (0.28) | -1.57 (0.21)
  Week 24 (N = 100, 105) | -2.00 (0.29) | -1.64 (0.23)
  Week 32 (N = 100, 105) | -1.78 (0.28) | -1.69 (0.23)
  Week 40 (N = 100, 105) | -2.12 (0.29) | -1.82 (0.24)
  Week 48 (N = 100, 105) | -2.17 (0.29) | -1.83 (0.25)
  Week 56 (N = 100, 105) | -2.13 (0.28) | -2.09 (0.25)
  Week 68 (N = 100, 105) | -2.15 (0.27) | -1.92 (0.25)
  Week 80 (N = 100, 105) | -2.18 (0.28) | -1.99 (0.26)
  Week 92 (N = 100, 105) | -2.33 (0.30) | -2.04 (0.26)
  Week 104 (N = 100, 105) | -2.37 (0.31) | -2.16 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0173, ANCOVA; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.19 to -0.12]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1618, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.97 to 0.16]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0153, ANCOVA; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.25 to -0.13]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0866, ANCOVA; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.05 to 0.07]

15. Secondary Outcome: Mean Change From Baseline in BASFI Getting Out of an Arm-less Chair at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.94 (0.28) | -0.53 (0.27)
  Week 4 (N= 105, 108) | -1.44 (0.28) | -0.84 (0.27)
  Week 8 (N= 105, 108) | -1.54 (0.29) | -1.02 (0.27)
  Week 12 (N = 105, 108) | -1.79 (0.28) | -1.07 (0.27)
  Week 16 (N = 100, 105) | -2.04 (0.29) | -1.90 (0.23)
  Week 24 (N = 100, 105) | -2.20 (0.29) | -2.12 (0.23)
  Week 32 (N = 100, 105) | -2.04 (0.29) | -2.18 (0.25)
  Week 40 (N = 100, 105) | -2.40 (0.30) | -2.38 (0.25)
  Week 48 (N = 100, 105) | -2.40 (0.29) | -2.25 (0.26)
  Week 56 (N = 100, 105) | -2.27 (0.28) | -2.47 (0.25)
  Week 68 (N = 100, 105) | -2.45 (0.28) | -2.46 (0.25)
  Week 80 (N = 100, 105) | -2.52 (0.28) | -2.33 (0.25)
  Week 92 (N = 100, 105) | -2.60 (0.29) | -2.48 (0.25)
  Week 104 (N = 100, 105) | -2.65 (0.29) | -2.48 (0.25)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1413, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.95 to 0.14]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0284, ANCOVA; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.14 to -0.06]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0659, ANCOVA; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.07 to 0.03]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0098, ANCOVA; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.26 to -0.18]

16. Secondary Outcome: Mean Change From Baseline in BASFI Physically Demanding Activities at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 104, 107) | -0.88 (0.26) | -0.13 (0.25)
  Week 4 (N= 104, 108) | -1.06 (0.28) | -0.26 (0.27)
  Week 8 (N= 104, 108) | -1.51 (0.28) | -0.80 (0.26)
  Week 12 (N = 104, 109) | -1.69 (0.29) | -0.91 (0.27)
  Week 16 (N = 99, 105) | -2.12 (0.26) | -1.79 (0.25)
  Week 24 (N = 99, 105) | -2.23 (0.26) | -2.05 (0.26)
  Week 32 (N = 99, 105) | -2.20 (0.25) | -2.19 (0.24)
  Week 40 (N = 99, 105) | -2.79 (0.26) | -2.24 (0.27)
  Week 48 (N = 99, 105) | -2.71 (0.27) | -2.25 (0.26)
  Week 56 (N = 99, 105) | -2.66 (0.27) | -2.37 (0.28)
  Week 68 (N = 99, 105) | -2.67 (0.26) | -2.60 (0.29)
  Week 80 (N = 99, 105) | -2.70 (0.26) | -2.39 (0.28)
  Week 92 (N = 99, 105) | -2.91 (0.27) | -2.59 (0.28)
  Week 104 (N = 99, 105) | -3.02 (0.27) | -2.59 (0.30)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0037, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.26 to -0.25]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0044, ANCOVA; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.35 to -0.25]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0104, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.26 to -0.17]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0060, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.33 to -0.22]

17. Secondary Outcome: Mean Change From Baseline in BASFI Reaching up High at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.33 (0.26) | -0.02 (0.24)
  Week 4 (N= 105, 108) | -0.63 (0.27) | -0.21 (0.26)
  Week 8 (N= 105, 108) | -0.81 (0.26) | -0.31 (0.25)
  Week 12 (N = 105, 109) | -0.70 (0.27) | -0.20 (0.25)
  Week 16 (N = 100, 105) | -1.09 (0.26) | -1.34 (0.22)
  Week 24 (N = 100, 105) | -1.26 (0.26) | -1.46 (0.22)
  Week 32 (N = 100, 105) | -1.00 (0.27) | -1.46 (0.23)
  Week 40 (N = 100, 105) | -1.30 (0.25) | -1.66 (0.24)
  Week 48 (N = 100, 105) | -1.38 (0.26) | -1.67 (0.25)
  Week 56 (N = 100, 105) | -1.34 (0.25) | -1.76 (0.24)
  Week 68 (N = 100, 105) | -1.42 (0.24) | -1.77 (0.24)
  Week 80 (N = 100, 105) | -1.37 (0.24) | -1.63 (0.24)
  Week 92 (N = 100, 105) | -1.55 (0.25) | -1.83 (0.24)
  Week 104 (N = 100, 105) | -1.62 (0.25) | -1.76 (0.24)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2268, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.80 to 0.19]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1145, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.93 to 0.10]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0512, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0509, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.02 to 0.00]

18. Secondary Outcome: Mean Change From Baseline in BASFI Climbing Steps Without Aid at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.46 (0.26) | -0.16 (0.24)
  Week 4 (N= 105, 108) | -0.65 (0.28) | -0.09 (0.26)
  Week 8 (N= 105, 108) | -0.92 (0.28) | -0.44 (0.27)
  Week 12 (N = 105, 109) | -0.93 (0.29) | -0.58 (0.27)
  Week 16 (N = 100, 105) | -1.48 (0.28) | -1.64 (0.24)
  Week 24 (N = 100, 105) | -1.54 (0.27) | -1.65 (0.25)
  Week 32 (N = 100, 105) | -1.57 (0.28) | -1.97 (0.25)
  Week 40 (N = 100, 105) | -1.84 (0.28) | -2.19 (0.26)
  Week 48 (N = 100, 105) | -1.78 (0.28) | -2.05 (0.28)
  Week 56 (N = 100, 105) | -1.81 (0.27) | -2.26 (0.26)
  Week 68 (N = 100, 105) | -1.88 (0.28) | -2.34 (0.28)
  Week 80 (N = 100, 105) | -1.89 (0.28) | -2.16 (0.26)
  Week 92 (N = 100, 105) | -1.91 (0.29) | -2.38 (0.28)
  Week 104 (N = 100, 105) | -2.01 (0.29) | -2.42 (0.28)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2430, ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.79 to 0.20]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0384, ANCOVA; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.09 to -0.03]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0797, ANCOVA; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.03 to 0.06]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2186, ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.90 to 0.21]

19. Secondary Outcome: Mean Change From Baseline in BASFI Getting-up Off-floor From Back at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.95 (0.28) | -0.53 (0.27)
  Week 8 (N= 105, 108) | -1.10 (0.28) | -0.77 (0.27)
  Week 12 (N = 105, 109) | -1.58 (0.31) | -1.18 (0.29)
  Week 12 (N= 105, 108) | -1.34 (0.30) | -1.05 (0.28)
  Week 16 (N = 100, 105) | -1.97 (0.28) | -2.18 (0.26)
  Week 24 (N = 100, 105) | -2.07 (0.26) | -2.18 (0.25)
  Week 32 (N = 100, 105) | -2.05 (0.27) | -2.31 (0.27)
  Week 40 (N = 100, 105) | -2.52 (0.27) | -2.59 (0.27)
  Week 48 (N = 100, 105) | -2.40 (0.28) | -2.51 (0.27)
  Week 56 (N = 100, 105) | -2.48 (0.27) | -2.81 (0.27)
  Week 68 (N = 100, 105) | -2.50 (0.27) | -2.75 (0.28)
  Week 80 (N = 100, 105) | -2.50 (0.26) | -2.63 (0.27)
  Week 92 (N = 100, 105) | -2.55 (0.29) | -2.84 (0.28)
  Week 104 (N = 100, 105) | -2.71 (0.29) | -2.90 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1410, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.96 to 0.14]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2299, ANCOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.88 to 0.21]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.3221, ANCOVA; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.87 to 0.29]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1891, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.99 to 0.20]

20. Secondary Outcome: Mean Change From Baseline in BASFI Standing Unsupported for 10 Minutes at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.58 (0.26) | -0.17 (0.24)
  Week 4 (N= 105, 108) | -0.80 (0.27) | -0.25 (0.25)
  Week 8 (N= 105, 108) | -1.03 (0.28) | -0.60 (0.27)
  Week 12 (N = 105, 109) | -1.33 (0.30) | -0.97 (0.29)
  Week 16 (N = 100, 105) | -1.88 (0.26) | -1.93 (0.23)
  Week 24 (N = 100, 105) | -1.96 (0.26) | -1.98 (0.25)
  Week 32 (N = 100, 105) | -1.84 (0.26) | -2.19 (0.25)
  Week 40 (N = 100, 105) | -2.17 (0.27) | -2.44 (0.26)
  Week 48 (N = 100, 105) | -2.30 (0.28) | -2.41 (0.28)
  Week 56 (N = 100, 105) | -2.26 (0.25) | -2.63 (0.26)
  Week 68 (N = 100, 105) | -2.37 (0.27) | -2.64 (0.27)
  Week 80 (N = 100, 105) | -2.41 (0.26) | -2.56 (0.26)
  Week 92 (N = 100, 105) | -2.42 (0.27) | -2.72 (0.28)
  Week 104 (N = 100, 105) | -2.53 (0.27) | -2.74 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1080, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.90 to 0.09]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0389, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.06 to -0.03]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1181, ANCOVA; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.98 to 0.11]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2271, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.94 to 0.22]

21. Secondary Outcome: Mean Change From Baseline in BASFI Looking Over Shoulder at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 8 (N= 105, 108) | -1.21 (0.28) | -0.84 (0.26)
  Week 12 (N = 105, 108) | -1.40 (0.28) | -0.82 (0.27)
  Week 16 (N = 100, 105) | -1.63 (0.28) | -1.69 (0.26)
  Week 24 (N = 100, 105) | -1.59 (0.28) | -1.84 (0.27)
  Week 32 (N = 100, 105) | -1.61 (0.29) | -1.92 (0.26)
  Week 40 (N = 100, 105) | -1.91 (0.28) | -2.03 (0.27)
  Week 48 (N = 100, 105) | -1.97 (0.28) | -2.08 (0.27)
  Week 56 (N = 100, 105) | -1.99 (0.27) | -2.27 (0.26)
  Week 68 (N = 100, 105) | -2.05 (0.27) | -2.25 (0.27)
  Week 80 (N = 100, 105) | -2.03 (0.27) | -1.94 (0.29)
  Week 92 (N = 100, 105) | -1.97 (0.28) | -2.19 (0.27)
  Week 104 (N = 100, 105) | -2.14 (0.27) | -2.16 (0.28)
  Week 2 (N= 105, 107) | -0.83 (0.27) | -0.07 (0.25)
  Week 4 (N= 105, 108) | -0.88 (0.28) | -0.33 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0044, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.27 to -0.24]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0455, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.09 to -0.01]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1750, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.91 to 0.17]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0379, ANCOVA; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.12 to -0.03]

22. Secondary Outcome: Mean Change From Baseline in BASFI Putting on Socks at Time Points
Description: as for outcome 12
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.94 (0.27) | -0.47 (0.26)
  Week 4 (N= 105, 108) | -0.74 (0.29) | -0.34 (0.27)
  Week 8 (N= 105, 108) | -1.04 (0.28) | -0.54 (0.27)
  Week 12 (N = 105, 108) | -1.02 (0.28) | -0.57 (0.26)
  Week 16 (N = 100, 105) | -1.52 (0.29) | -1.36 (0.21)
  Week 24 (N = 100, 105) | -1.65 (0.29) | -1.44 (0.21)
  Week 32 (N = 100, 105) | -1.55 (0.29) | -1.49 (0.21)
  Week 40 (N = 100, 105) | -1.92 (0.28) | -1.64 (0.23)
  Week 48 (N = 100, 105) | -1.95 (0.28) | -1.60 (0.23)
  Week 56 (N = 100, 105) | -1.85 (0.29) | -1.75 (0.21)
  Week 68 (N = 100, 105) | -1.80 (0.27) | -1.62 (0.22)
  Week 80 (N = 100, 105) | -1.92 (0.29) | -1.66 (0.22)
  Week 92 (N = 100, 105) | -1.93 (0.29) | -1.70 (0.22)
  Week 104 (N = 100, 105) | -1.95 (0.29) | -1.71 (0.23)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0826, ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.98 to 0.06]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1538, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.96 to 0.15]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0728, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.04 to 0.05]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0975, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.99 to 0.08]

23. Secondary Outcome: Changes From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Time Points
Description: BASDAI is a validated self assessment tool used to determine disease activity in participant with Ankylosing Spondylitis (AS). Utilizing a VAS of 0-10 (0 = none and 10 = very severe) participant's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI score is obtained by computing the mean score for the 2 questions related to morning stiffness (questions 5 and 6) and then adding that value to the sum of the scores for the first 4 questions and then dividing the total by 5. This can be written as BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5. The final BASDAI score averages the individual assessments for a final score range of 0-10.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N = 105, 108) | -0.96 (0.23) | -0.39 (0.22)
  Week 4 (N = 105, 109) | -1.63 (0.24) | -0.97 (0.22)
  Week 8 (N = 105, 109) | -2.05 (0.26) | -1.24 (0.25)
  Week 12 (N = 105, 109) | -1.96 (0.28) | -1.31 (0.27)
  Week 16 (N = 100, 105) | -2.70 (0.21) | -2.98 (0.20)
  Week 24 (N = 100, 105) | -2.86 (0.22) | -3.26 (0.19)
  Week 32 (N = 100, 105) | -2.72 (0.22) | -3.24 (0.22)
  Week 40 (N = 100, 105) | -3.22 (0.22) | -3.41 (0.21)
  Week 48 (N = 100, 105) | -3.18 (0.23) | -3.47 (0.22)
  Week 56 (N = 100, 105) | -3.21 (0.24) | -3.50 (0.21)
  Week 68 (N = 100, 105) | -3.17 (0.23) | -3.69 (0.22)
  Week 80 (N = 100, 105) | -3.12 (0.24) | -3.59 (0.22)
  Week 92 (N = 100, 105) | -3.35 (0.25) | -3.77 (0.23)
  Week 104 (N = 100, 105) | -3.41 (0.24) | -3.87 (0.23)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0186, ANCOVA; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.18 to -0.11]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0106, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.01 to -0.13]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0048, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.11 to -0.20]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.31 to -0.31]

24. Secondary Outcome: Mean Change From Baseline in BASDAI Level of Morning Stiffness at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | -1.26 (0.29) | -0.45 (0.28)
  Week 4 (N= 105, 108) | -1.83 (0.31) | -1.00 (0.29)
  Week 8 (N= 101, 106) | -2.46 (0.33) | -1.24 (0.31)
  Week 12 (N = 101, 106) | -2.26 (0.34) | -1.43 (0.32)
  Week 16 (N = 100, 105) | -3.50 (0.29) | -3.40 (0.25)
  Week 24 (N = 100, 105) | -3.71 (0.28) | -4.00 (0.25)
  Week 32 (N = 100, 105) | -3.45 (0.28) | -3.84 (0.26)
  Week 40 (N = 100, 105) | -3.93 (0.28) | -4.23 (0.24)
  Week 48 (N = 100, 105) | -3.91 (0.30) | -4.06 (0.25)
  Week 56 (N = 100, 105) | -3.89 (0.31) | -4.28 (0.25)
  Week 68 (N = 100, 105) | -3.99 (0.28) | -4.41 (0.26)
  Week 80 (N = 100, 105) | -3.74 (0.29) | -4.30 (0.26)
  Week 92 (N = 100, 105) | -3.99 (0.31) | -4.42 (0.25)
  Week 104 (N = 100, 105) | -4.09 (0.30) | -4.66 (0.24)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0058, ANCOVA; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.37 to -0.24]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0064, ANCOVA; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.42 to -0.24]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.85 to -0.60]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0134, ANCOVA; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.49 to -0.17]

25. Secondary Outcome: Mean Change From Baseline in BASDAI Level of Fatigue/Tiredness at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | -0.80 (0.27) | -0.23 (0.26)
  Week 4 (N= 105, 109) | -1.71 (0.28) | -1.26 (0.26)
  Week 8 (N= 105, 109) | -1.98 (0.30) | -1.29 (0.29)
  Week 12 (N = 105, 109) | -1.70 (0.34) | -1.32 (0.32)
  Week 16 (N = 100, 105) | -2.29 (0.24) | -2.89 (0.25)
  Week 24 (N = 100, 105) | -2.48 (0.27) | -2.95 (0.23)
  Week 32 (N = 100, 105) | -2.22 (0.26) | -2.74 (0.26)
  Week 40 (N = 100, 105) | -2.82 (0.26) | -2.93 (0.26)
  Week 48 (N = 100, 105) | -2.86 (0.25) | -3.19 (0.26)
  Week 56 (N = 100, 105) | -3.03 (0.26) | -3.20 (0.26)
  Week 68 (N = 100, 105) | -2.92 (0.27) | -3.48 (0.24)
  Week 80 (N = 100, 105) | -3.15 (0.28) | -3.36 (0.26)
  Week 92 (N = 100, 105) | -3.20 (0.27) | -3.68 (0.25)
  Week 104 (N = 100, 105) | -3.18 (0.27) | -3.63 (0.28)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0316, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.09 to -0.05]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0973, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.99 to 0.08]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0216, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.27 to -0.10]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2425, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.03 to 0.26]

26. Secondary Outcome: Mean Change From Baseline in BASDAI Level of Discomfort at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | -0.81 (0.31) | -0.48 (0.29)
  Week 8 (N= 105, 109) | -1.31 (0.33) | -0.77 (0.31)
  Week 12 (N= 105, 109) | -1.91 (0.33) | -1.20 (0.31)
  Week 12 (N = 105, 109) | -1.68 (0.34) | -1.29 (0.32)
  Week 16 (N = 100, 105) | -2.65 (0.30) | -2.82 (0.25)
  Week 24 (N = 100, 105) | -2.71 (0.31) | -3.07 (0.26)
  Week 32 (N = 100, 105) | -2.64 (0.31) | -3.25 (0.27)
  Week 40 (N = 100, 105) | -3.09 (0.30) | -3.25 (0.27)
  Week 48 (N = 100, 105) | -2.97 (0.33) | -3.27 (0.29)
  Week 56 (N = 100, 105) | -3.13 (0.34) | -3.24 (0.29)
  Week 68 (N = 100, 105) | -3.01 (0.32) | -3.49 (0.31)
  Week 80 (N = 100, 105) | -2.87 (0.33) | -3.50 (0.28)
  Week 92 (N = 100, 105) | -3.21 (0.33) | -3.57 (0.30)
  Week 104 (N = 100, 105) | -3.31 (0.34) | -3.72 (0.29)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2688, ANCOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.92 to 0.26]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0866, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.17 to 0.08]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0277, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.34 to -0.08]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2390, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.04 to 0.26]

27. Secondary Outcome: Mean Change From Baseline in BASDAI Level of How Long Stiffness Lasts at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | -0.61 (0.28) | -0.15 (0.26)
  Week 4 (N= 105, 109) | -1.33 (0.29) | -0.62 (0.28)
  Week 8 (N= 105, 109) | -1.62 (0.30) | -0.68 (0.29)
  Week 12 (N = 105, 109) | -1.98 (0.31) | -0.97 (0.29)
  Week 16 (N = 100, 105) | -2.63 (0.27) | -2.60 (0.26)
  Week 24 (N = 100, 105) | -2.84 (0.29) | -3.04 (0.29)
  Week 32 (N = 100, 105) | -2.54 (0.29) | -3.06 (0.30)
  Week 40 (N = 100, 105) | -2.94 (0.30) | -3.28 (0.30)
  Week 48 (N = 100, 105) | -2.90 (0.30) | -3.09 (0.32)
  Week 56 (N = 100, 105) | -2.92 (0.33) | -3.17 (0.30)
  Week 68 (N = 100, 105) | -2.91 (0.32) | -3.50 (0.32)
  Week 80 (N = 100, 105) | -2.77 (0.30) | -3.24 (0.31)
  Week 92 (N = 100, 105) | -2.89 (0.33) | -3.36 (0.31)
  Week 104 (N = 100, 105) | -2.95 (0.32) | -3.38 (0.31)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0928, ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-1.00 to 0.08]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0139, ANCOVA; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.27 to -0.15]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0017, ANCOVA; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.53 to -0.36]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.61 to -0.43]

28. Secondary Outcome: Mean Change From Baseline in BASDAI Level of Pain/Swelling at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 107) | -0.64 (0.32) | -0.41 (0.30)
  Week 4 (N= 105, 109) | -1.35 (0.32) | -0.68 (0.31)
  Week 8 (N= 105, 109) | -1.69 (0.33) | -1.01 (0.31)
  Week 12 (N = 105, 109) | -1.47 (0.33) | -0.87 (0.32)
  Week 16 (N = 100, 105) | -2.38 (0.28) | -2.66 (0.28)
  Week 24 (N = 100, 105) | -2.49 (0.29) | -2.92 (0.28)
  Week 32 (N = 100, 105) | -2.47 (0.30) | -3.10 (0.29)
  Week 40 (N = 100, 105) | 2.91 (0.27) | -3.21 (0.28)
  Week 48 (N = 100, 105) | -2.80 (0.30) | -3.21 (0.30)
  Week 56 (N = 100, 105) | -2.66 (0.31) | -3.13 (0.29)
  Week 68 (N = 100, 105) | -2.60 (0.32) | -3.24 (0.32)
  Week 80 (N = 100, 105) | -2.67 (0.32) | -3.19 (0.31)
  Week 92 (N = 100, 105) | -2.96 (0.31) | -3.40 (0.32)
  Week 104 (N = 100, 105) | -3.07 (0.31) | -3.51 (0.31)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4559, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.84 to 0.38]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0345, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.28 to -0.05]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0340, ANCOVA; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.30 to -0.05]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0634, ANCOVA; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.24 to 0.03]

29. Secondary Outcome: Mean Change From Baseline in BASDAI Level of Neck/Back/Hip Pain at Time Points
Description: as for outcome 23
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | -1.34 (0.29) | -0.34 (0.28)
  Week 4 (N= 105, 109) | -1.91 (0.31) | -1.10 (0.29)
  Week 8 (N= 105, 109) | -2.32 (0.33) | -1.48 (0.31)
  Week 12 (N = 105, 109) | -2.44 (0.35) | -1.58 (0.33)
  Week 16 (N = 100, 105) | -3.13 (0.28) | -3.55 (0.28)
  Week 24 (N = 100, 105) | -3.32 (0.27) | -3.82 (0.26)
  Week 32 (N = 100, 105) | -3.27 (0.26) | -3.65 (0.27)
  Week 40 (N = 100, 105) | -3.81 (0.27) | -3.92 (0.27)
  Week 48 (N = 100, 105) | -3.85 (0.27) | -4.10 (0.26)
  Week 56 (N = 100, 105) | -3.82 (0.27) | -4.22 (0.27)
  Week 68 (N = 100, 105) | -3.83 (0.26) | -4.28 (0.27)
  Week 80 (N = 100, 105) | -3.60 (0.28) | -4.11 (0.28)
  Week 92 (N = 100, 105) | -3.88 (0.29) | -4.29 (0.28)
  Week 104 (N = 100, 105) | -3.96 (0.29) | -4.48 (0.27)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0007, ANCOVA; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.56 to -0.43]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0073, ANCOVA; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.39 to -0.22]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0094, ANCOVA; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-1.48 to -0.21]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0120, ANCOVA; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.54 to -0.19]

30. Secondary Outcome: Percentage of Participants With BASDAI 50 at Time Points
Description: Response was defined as a 50% improvement of the Baseline BASDAI to 104 weeks of study treatment, respectively. The BASDAI score is obtained by computing the mean score for the 2 questions related to morning stiffness (questions 5 and 6) and then adding that value to the sum of the scores for the first 4 questions and then dividing the total by 5. This can be written as BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
Percentage of participants
  Week 2 (N = 105, 108) | 17.14 | 5.56
  Week 4 (N = 105, 109) | 24.76 | 11.01
  Week 8 (N = 105, 109) | 37.14 | 22.02
  Week 12 (N = 105, 109) | 43.81 | 23.85
  Week 16 (N = 100, 105) | 45.00 | 59.05
  Week 24 (N = 100, 105) | 50.00 | 62.86
  Week 32 (N = 100, 105) | 49.00 | 59.05
  Week 40 (N = 100, 105) | 58.00 | 61.90
  Week 48 (N = 100, 105) | 60.00 | 64.76
  Week 56 (N = 100, 105) | 59.00 | 65.71
  Week 68 (N = 100, 105) | 61.00 | 66.67
  Week 80 (N = 100, 105) | 56.00 | 66.67
  Week 92 (N = 100, 105) | 62.00 | 71.43
  Week 104 (N = 100, 105) | 64.00 | 70.48
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0029, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 19.96, 95% CI 2-sided [7.54 to 32.37]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0100, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 11.59, 95% CI 2-sided [3.18 to 19.99]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0120, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.75, 95% CI 2-sided [3.62 to 23.89]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0213, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.12, 95% CI 2-sided [3.04 to 27.20]

31. Secondary Outcome: Percentage of Participants With BASDAI 20 at Time Points
Description: Response was defined as a 20% improvement of the Baseline BASDAI to 104 weeks of study treatment. The BASDAI score is obtained by computing the mean score for the 2 questions related to morning stiffness (questions 5 and 6) and then adding that value to the sum of the scores for the first 4 questions and then dividing the total by 5. This can be written as BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 109
Percentage of participants
  Week 2 (N = 105, 108) | 41.90 | 33.33
  Week 4 (N = 105, 109) | 56.19 | 42.20
  Week 8 (N = 105, 109) | 66.67 | 51.38
  Week 12 (N = 105, 109) | 64.76 | 56.88
  Week 16 (N = 100, 105) | 73.00 | 82.86
  Week 24 (N = 100, 105) | 77.00 | 86.67
  Week 32 (N = 100, 105) | 77.00 | 84.76
  Week 40 (N = 100, 105) | 86.00 | 87.62
  Week 48 (N = 100, 105) | 81.00 | 87.62
  Week 56 (N = 100, 105) | 81.00 | 85.71
  Week 68 (N = 100, 105) | 80.00 | 90.48
  Week 80 (N = 100, 105) | 81.00 | 88.57
  Week 92 (N = 100, 105) | 82.00 | 88.57
  Week 104 (N = 100, 105) | 84.00 | 90.48
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2755, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 7.88, 95% CI 2-sided [-5.15 to 20.92]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1950, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 8.57, 95% CI 2-sided [-4.39 to 21.54]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0278, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 13.99, 95% CI 2-sided [0.72 to 27.26]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0174, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 15.29, 95% CI 2-sided [2.28 to 28.30]

32. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Total Score at Time Points
Description: The BAS-G was a 2 question assessment evaluating the effect of AS on the participants well-being over the last week and last 6 months. The 2 questions were: How have you been over the last week? and How have you been over the last six months?. Each question is scored by the participant on a 100 mm scale ranging from 0 (Very Good) to 100 (Very Bad). The two values are averaged to obtain the BAS-G score.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 4 (N = 105, 109) | -1.29 (0.24) | -0.75 (0.22)
  Week 12 (N = 105, 109) | -1.85 (0.27) | -1.35 (0.25)
  Week 24 (N = 100, 105) | -2.80 (0.24) | -2.87 (0.19)
  Week 48 (N = 105, 109) | -3.20 (0.25) | -3.51 (0.22)
  Week 68 (N = 105, 109) | -3.28 (0.25) | -3.77 (0.23)
  Week 92 (N = 105, 109) | -3.55 (0.25) | -3.81 (0.23)
  Week 104 (N = 105, 109) | -3.59 (0.26) | -3.92 (0.24)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4 and 12 data only. Week 4; Test type: Superiority or Other; p = 0.0201, ANCOVA; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.99 to -0.09]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4 and 12 data only. Week 12; Test type: Superiority or Other; p = 0.0558, ANCOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.02 to 0.01]

33. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) Total Score at Time Points
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 104 | 109
Units on a scale
  Week 2 (N = 103, 108) | -0.08 (0.12) | -0.13 (0.11)
  Week 4 (N = 103, 109) | -0.30 (0.12) | -0.20 (0.11)
  Week 8 (N = 103, 109) | -0.36 (0.14) | -0.41 (0.13)
  Week 12 (N = 103, 109) | -0.34 (0.14) | -0.19 (0.10)
  Week 16 (N = 98, 105) | -0.44 (0.14) | -0.35 (0.10)
  Week 24 (N = 98, 105) | -0.48 (0.13) | -0.34 (0.10)
  Week 40 (N = 98, 105) | -0.49 (0.14) | -0.49 (0.11)
  Week 32 (N = 98, 105) | -0.55 (0.14) | -0.47 (0.11)
  Week 48 (N = 98, 105) | -0.54 (0.13) | -0.44 (0.11)
  Week 56 (N = 98, 105) | -0.56 (0.13) | -0.49 (0.11)
  Week 68 (N = 98, 105) | -0.60 (0.13) | -0.58 (0.11)
  Week 80 (N = 98, 105) | -0.64 (0.14) | -0.62 (0.11)
  Week 92 (N = 98, 105) | -0.61 (0.13) | -0.62 (0.11)
  Week 104 (N = 98, 105) | -0.61 (0.14) | -0.55 (0.11)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test, after Week 24. For label period results include unadjusted mean changes and standard errors, no covariate adjustments were applied; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6741, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.18 to 0.28]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3896, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.33 to 0.13]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.7468, ANCOVA; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.22 to 0.31]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.6871, ANCOVA; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.35 to 0.23]

34. Secondary Outcome: Mean Change From Baseline in BASMI Lateral Side Flexion Score by Time Point
Description: as for outcome 33
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 104 | 109
Units on a scale
  Week 2 (N= 100, 105) | 1.06 (0.49) | 0.69 (0.46)
  Week 4 (N= 100, 106) | 1.49 (0.51) | 1.49 (0.48)
  Week 8 (N= 100, 106) | 1.64 (0.53) | 0.91 (0.50)
  Week 12 (N = 100, 106) | 1.64 (0.62) | 0.43 (0.58)
  Week 16 (N = 98, 105) | 1.35 (0.55) | 1.02 (0.32)
  Week 24 (N = 98, 105) | 1.97 (0.66) | 1.29 (0.34)
  Week 32 (N = 98, 105) | 2.03 (0.57) | 1.62 (0.35)
  Week 40 (N = 98, 105) | 1.86 (0.59) | 1.57 (0.38)
  Week 48 (N = 98, 105) | 2.20 (0.55) | 1.36 (0.34)
  Week 56 (N = 98, 105) | 1.82 (0.54) | 1.43 (0.36)
  Week 68 (N = 98, 105) | 2.24 (0.58) | 1.54 (0.41)
  Week 80 (N = 98, 105) | 1.96 (0.59) | 1.52 (0.40)
  Week 92 (N = 98, 105) | 2.14 (0.60) | 1.50 (0.38)
  Week 104 (N = 98, 105) | 1.97 (0.59) | 1.65 (0.37)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4332, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.57 to 1.32]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.9947, ANCOVA; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.98 to 0.98]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1558, ANCOVA; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-0.28 to 1.75]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0488, ANCOVA; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [0.03 to 2.39]

35. Secondary Outcome: Mean Change From Baseline in BASMI Cervical Rotation Degree by Time Point
Description: as for outcome 33
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 109
Units on a scale
  Week 2 (N= 105, 108) | 1.35 (1.26) | 0.98 (1.19)
  Week 4 (N= 105, 109) | 3.52 (1.31) | 2.49 (1.23)
  Week 8 (N= 105, 109) | 4.92 (1.42) | 3.86 (1.34)
  Week 12 (N = 105, 109) | 4.46 (1.52) | 2.07 (1.44)
  Week 16 (N = 100, 105) | 5.13 (1.37) | 4.73 (1.09)
  Week 24 (N = 100, 105) | 5.00 (1.35) | 5.10 (1.18)
  Week 32 (N = 100, 105) | 5.32 (1.43) | 6.00 (1.25)
  Week 40 (N = 100, 105) | 5.56 (1.51) | 5.61 (1.19)
  Week 48 (N = 100, 105) | 5.04 (1.48) | 6.90 (1.19)
  Week 56 (N = 100, 105) | 5.70 (1.44) | 6.92 (1.31)
  Week 68 (N = 100, 105) | 6.47 (1.43) | 8.10 (1.23)
  Week 80 (N = 100, 105) | 6.14 (1.45) | 7.96 (1.23)
  Week 92 (N = 100, 105) | 6.26 (1.50) | 8.25 (1.24)
  Week 104 (N = 100, 105) | 5.92 (1.57) | 8.55 (1.22)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7645, ANCOVA; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-2.06 to 2.80]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4178, ANCOVA; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [-1.48 to 3.55]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.4430, ANCOVA; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-1.67 to 3.79]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.1095, ANCOVA; Mean Difference (Final Values) = 2.39, 95% CI 2-sided [-0.54 to 5.31]

36. Secondary Outcome: Mean Change From Baseline in BASMI Modified Schobers Test Score by Time Point
Description: as for outcome 33
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 104 | 109
Units on a scale
  Week 2 (N= 89, 90) | 0.17 (0.24) | 0.16 (0.23)
  Week 4 (N= 89, 90) | 0.02 (0.26) | 0.20 (0.25)
  Week 8 (N= 89, 90) | 0.15 (0.26) | 0.12 (0.25)
  Week 12 (N = 89, 90) | 0.05 (0.31) | 0.04 (0.30)
  Week 16 (N = 86, 86) | 0.71 (0.23) | 0.37 (0.24)
  Week 24 (N = 86, 86) | 0.98 (0.27) | 0.54 (0.25)
  Week 32 (N = 86, 86) | 0.73 (0.30) | 0.54 (0.28)
  Week 40 (N = 86, 86) | 0.68 (0.24) | 0.77 (0.25)
  Week 48 (N = 86, 86) | 0.75 (0.26) | 0.63 (0.26)
  Week 56 (N = 86, 86) | 1.16 (0.36) | 0.79 (0.32)
  Week 68 (N = 86, 86) | 1.34 (0.35) | 0.89 (0.31)
  Week 80 (N = 86, 86) | 1.38 (0.38) | 0.97 (0.31)
  Week 92 (N = 86, 86) | 1.03 (0.35) | 0.88 (0.29)
  Week 104 (N = 86, 86) | 0.99 (0.36) | 0.92 (0.33)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9504, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.46 to 0.49]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4971, ANCOVA; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.70 to 0.34]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.8999, ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.47 to 0.54]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.9712, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.60 to 0.62]

37. Secondary Outcome: Mean Change From Baseline in BASMI Intermalleolar Distance Score by Time Point
Description: as for outcome 33
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 104 | 109
Units on a scale
  Week 2 (N= 105, 108) | 0.75 (1.22) | -0.15 (1.15)
  Week 4 (N= 105, 109) | 4.02 (1.50) | 1.17 (1.42)
  Week 8 (N= 105, 109) | 4.25 (1.70) | 1.99 (1.61)
  Week 12 (N = 105, 109) | 3.25 (1.75) | 1.81 (1.66)
  Week 16 (N = 100, 105) | 6.28 (1.44) | 3.73 (1.27)
  Week 24 (N = 100, 105) | 7.48 (1.41) | 4.76 (1.30)
  Week 32 (N = 100, 105) | 8.09 (1.38) | 5.01 (1.35)
  Week 40 (N = 100, 105) | 8.38 (1.38) | 5.61 (1.34)
  Week 48 (N = 100, 105) | 8.35 (1.50) | 6.32 (1.33)
  Week 56 (N = 100, 105) | 9.31 (1.48) | 7.42 (1.38)
  Week 68 (N = 100, 105) | 9.26 (1.55) | 7.92 (1.37)
  Week 80 (N = 100, 105) | 9.17 (1.55) | 8.73 (1.32)
  Week 92 (N = 100, 105) | 9.80 (1.55) | 9.05 (1.34)
  Week 104 (N = 100, 105) | 8.91 (1.57) | 8.72 (1.35)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4556, ANCOVA; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-1.46 to 3.24]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0543, ANCOVA; Mean Difference (Final Values) = 2.85, 95% CI 2-sided [-0.05 to 5.75]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1754, ANCOVA; Mean Difference (Final Values) = 2.26, 95% CI 2-sided [-1.02 to 5.53]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.3985, ANCOVA; Mean Difference (Final Values) = 1.45, 95% CI 2-sided [-1.93 to 4.82]

38. Secondary Outcome: Mean Change From Baseline in BASMI Tragus to Wall Score by Time Point
Description: as for outcome 33
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 104 | 109
Units on a scale
  Week 2 (N= 105, 108) | 0.02 (0.21) | -0.20 (0.20)
  Week 4 (N= 105, 109) | -0.20 (0.21) | -0.37 (0.20)
  Week 8 (N= 105, 109) | -0.31 (0.20) | -0.44 (0.19)
  Week 12 (N = 105, 109) | -0.29 (0.23) | -0.41 (0.22)
  Week 16 (N = 100, 105) | 0.14 (0.22) | -0.02 (0.16)
  Week 24 (N = 100, 105) | 0.28 (0.24) | 0.01 (0.17)
  Week 32 (N = 100, 105) | 0.02 (0.27) | 0.01 (0.16)
  Week 40 (N = 100, 105) | -0.07 (0.25) | -0.08 (0.21)
  Week 48 (N = 100, 105) | -0.16 (0.27) | 0.03 (0.16)
  Week 68 (N = 100, 105) | -0.28 (0.27) | 0.08 (0.18)
  Week 56 (N = 100, 105) | 0.01 (0.26) | -0.00 (0.17)
  Week 80 (N = 100, 105) | -0.24 (0.26) | -0.00 (0.16)
  Week 92 (N = 100, 105) | -0.17 (0.27) | -0.02 (0.18)
  Week 104 (N = 100, 105) | -0.39 (0.25) | -0.15 (0.18)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2823, ANCOVA; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.18 to 0.62]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.4029, ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.23 to 0.58]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.5110, ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.25 to 0.51]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.5844, ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.32 to 0.56]

39. Secondary Outcome: Change From Baseline in Chest Expansion at Time Points
Description: Chest expansion, measured in cm, is defined as the difference in thoracic circumference during full expiration versus full inspiration, measured at the fourth intercostal space (nipple line). At maximal inspiration, the chest circumference was measured at nipple line or at the 4th intercostal space (in cm to the nearest 0.1 cm).
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
cm
  Week 2 (N = 104, 105) | 0.16 (0.22) | 0.69 (0.20)
  Week 4 (N = 104, 108) | 0.31 (0.25) | 0.44 (0.23)
  Week 8 (N = 104, 108) | 0.20 (0.25) | 0.61 (0.23)
  Week 12 (N = 104, 108) | 0.12 (0.25) | 0.37 (0.24)
  Week 16 (N = 99, 104) | 0.43 (0.19) | 0.68 (0.19)
  Week 24 (N = 99, 104) | 0.38 (0.17) | 0.69 (0.19)
  Week 32 (N = 99, 104) | 0.49 (0.18) | 0.62 (0.18)
  Week 40 (N = 99, 104) | 0.55 (0.17) | 0.71 (0.17)
  Week 48 (N = 99, 104) | 0.63 (0.17) | 0.80 (0.21)
  Week 56 (N = 99, 104) | 0.49 (0.18) | 0.72 (0.19)
  Week 68 (N = 99, 104) | 0.61 (0.17) | 0.56 (0.18)
  Week 80 (N = 99, 104) | 0.32 (0.18) | 0.74 (0.20)
  Week 92 (N = 99, 104) | 0.52 (0.18) | 0.56 (0.20)
  Week 104 (N = 99, 104) | 0.67 (0.18) | 0.63 (0.20)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Most within group comparisons to baseline were <0.001, from paired t-test. For open-label period results include unadjusted mean changes and standard errors, no covariate adjustments were applied; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0129, ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.95 to -0.11]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.6003, ANCOVA; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.61 to 0.35]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0911, ANCOVA; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.89 to 0.07]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.3144, ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.73 to 0.24]

40. Secondary Outcome: Mean Change From Baseline in Occiput-to-wall Test at Time Points
Description: Occiput-to-wall distance: distance between the occiput (posterior or back portion of the head) and the wall when the participant stood with heels and shoulder against the wall and the back straight.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: cm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
cm
  Week 2 (N = 104, 106) | -0.21 (0.19) | -0.12 (0.19)
  Week 4 (N = 104, 108) | -0.37 (0.20) | -0.36 (0.19)
  Week 8 (N = 104, 108) | -0.09 (0.24) | -0.27 (0.23)
  Week 12 (N = 104, 108) | -0.28 (0.24) | -0.41 (0.23)
  Week 16 (N = 99, 104) | -0.24 (0.25) | -0.29 (0.11)
  Week 24 (N = 99, 104) | -0.11 (0.25) | -0.38 (0.18)
  Week 32 (N = 99, 104) | -0.20 (0.25) | -0.31 (0.16)
  Week 40 (N = 99, 104) | -0.34 (0.22) | -0.24 (0.17)
  Week 48 (N = 99, 104) | -0.25 (0.24) | -0.42 (0.13)
  Week 56 (N = 99, 104) | -0.42 (0.22) | -0.26 (0.14)
  Week 68 (N = 99, 104) | -0.42 (0.23) | -0.21 (0.16)
  Week 80 (N = 99, 104) | -0.34 (0.24) | -0.55 (0.17)
  Week 92 (N = 99, 104) | -0.29 (0.24) | -0.49 (0.15)
  Week 104 (N = 99, 104) | -0.73 (0.26) | -0.52 (0.19)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 39, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12, data only. Week 2; Test type: Superiority or Other; p = 0.6476, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.46 to 0.29]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12, data only. Week 4; Test type: Superiority or Other; p = 0.9777, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.40 to 0.39]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12, data only. Week 8; Test type: Superiority or Other; p = 0.4453, ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.28 to 0.65]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12, data only. Week 12; Test type: Superiority or Other; p = 0.5782, ANCOVA; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.33 to 0.60]

41. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) - Spine 6 Discovertebral Units (DVU) Total Score at 12 Weeks
Description: The change from baseline in the MRI score of spine was assessed using SPARCC method. The scores of the 6 most severely affected spinal levels (discovertebral units/DVUs) was selected. Each DVU was divided into 4 quadrants. Each quadrant was assigned a score of 0 = no lesion or 1 = increased signal. This was repeated for each of 3 consecutive sagittal slices resulting in a score of up to 12 per DVU. On each slice, the presence of a lesion exhibiting an intense signal in any quadrant was assigned an additional score of 1 for that slice. Additionally, on each slice the presence of a lesion exhibiting depth ≥ 1 cm in any quadrant was given an additional score of 1. The maximum score for 6 DVU Spine Total Score is 108.
Time Frame: Week 12
Population: mITT population defined as all randomized participants who took at least one dose of study drug, had at least one on-therapy evaluation and met the ASAS classification criteria for AxSpA. Missing data were imputed through observed cases.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 95 | 105
units on a scale | -2.12 (0.72) | -2.12 (0.43)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0414, ANCOVA; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.88 to -0.04]

42. Secondary Outcome: Mean Change From Baseline in SPARCC Score for the Sacroiliac Joint at Time Points
Description: The change from baseline in the MRI score of sacroiliac joints was assessed using SPARCC method. Scoring was based on 6 consecutive coronal slices from posterior to anterior. Each joint was divided into 4 quadrants. Each quadrant was assigned a score of 0 = no lesion/1 = increased signal. For each slice, the score is increased by 1 for each joint that exhibits an intense signal in any quadrant. Also, for each slice, an additional score of 1 will be given for each joint that includes a lesion demonstrating continuous increased signal of a depth ≥1 cm from the articular surface. The maximum possible score is 72.
Time Frame: Weeks 12 and 104
Population: as for outcome 41
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 95 | 105
units on a scale
  Week 12 (N = 97, 105) | -3.99 (0.72) | -0.86 (0.43)
  Week 104 (N = 74, 79) | -6.00 (1.15) | -3.36 (0.84)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.93, 95% CI 2-sided [-4.16 to -1.70]

43. Secondary Outcome: Mean Change From Baseline in SPARCC - Spine 6 Discovertebral Units (DVU) Total Score at Time Points
Description: as for outcome 41
Time Frame: Weeks 12 and 104
Population: as for outcome 41
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 95 | 105
units on a scale
  Week 12 (N= 95, 105) | -2.12 (0.49) | -1.16 (0.47)
  Week 104 (N= 74, 80) | -2.08 (0.91) | -0.78 (0.49)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0414, ANCOVA; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.88 to -0.04]

44. Secondary Outcome: Mean Change From Baseline in Ankylosing Spondylitis Spine Magnetic Resonance Imaging-Activity (ASspiMRI-a) Total Score
Description: ASspiMRI-a measures acute lesion scores as determined by short-tau inversion recovery (STIR) and gadolinium-enhanced T1 (Gd-DTPA). All 23 disco-vertebral units (DVU) of the spine (from C2 to S1), defined as the region between 2 virtual lines through the middle of each vertebra, are scored in a single dimension, which is representing the highest level of inflammation in that particular DVU. Enhancement and bone marrow edema are graded (0-3) for each DVU, with 3 more grades (4-6) if, in addition to the signs of acute inflammation defined for grades 1-3, erosions are visualized, leading to a maximum score of 138 for the entire spine. Acute spinal changes were assessed by using STIR sagittal views of the cervical, thoracic and lumbar spine. The total score ranges from 0 (no inflammation) to 138 (high inflammation).
Time Frame: Weeks 12 and 104
Population: as for outcome 41
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 95 | 105
Units on a scale
  Week 12 (N= 95 105) | -0.73 (0.17) | -0.33 (0.16)
  Week 104 (N= 73, 80) | -0.79 (0.29) | -0.28 (0.16)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.0132, ANCOVA; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.72 to -0.08]

45. Secondary Outcome: Mean Change From Baseline in Number of Swollen Joints at Time Points
Description: Forty-four (44) joints were assessed by the Investigator to determine the number of joints that were considered swollen (artificial joints were not assessed). The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done. The 44 joints to be assessed were:sternoclavicular, acromioclavicular, shoulder, elbow, wrist (includes radiocarpal, carpal and carpometacarpal considered as one unit), metacarpophalangeals (I, II, III, IV, V), thumb interphalangeal (IP), proximal IPs (II, III, IV, V), knee, ankle, metatarsophalangeals (I, II, III, IV, V).
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of joints
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 102 | 105
Number of joints
  Week 2 (N = 100, 102) | -0.27 (0.17) | -0.08 (0.16)
  Week 4 (N = 100, 105) | -0.62 (0.13) | -0.45 (0.13)
  Week 8 (N = 101, 105) | -0.71 (0.14) | -0.52 (0.13)
  Week 12 (N = 101, 105) | -0.60 (0.12) | -0.29 (0.11)
  Week 16 (N = 96, 102) | -0.76 (0.17) | -0.59 (0.19)
  Week 24 (N = 96, 102) | -0.80 (0.20) | -0.68 (0.22)
  Week 32 (N= 96, 102) | -0.75 (0.23) | -0.64 (0.20)
  Week 40 (N= 96, 102) | -0.80 (0.21) | -0.71 (0.20)
  Week 48 (N= 96, 102) | -0.83 (0.21) | -0.83 (0.22)
  Week 56 (N= 96, 102) | -0.86 (0.21) | -0.76 (0.21)
  Week 68 (N= 96, 102) | -0.86 (0.21) | -0.82 (0.22)
  Week 80 (N= 96, 102) | -0.85 (0.21) | -0.79 (0.22)
  Week 92 (N= 96, 102) | -0.83 (0.21) | -0.76 (0.23)
  Week 104 (N= 96, 102) | -0.89 (0.21) | -0.84 (0.22)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2438, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.52 to 0.13]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1958, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.42 to 0.09]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1624, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.46 to 0.08]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0091, ANCOVA; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.54 to -0.08]

46. Secondary Outcome: Mean Change From Baseline in Number of Tender Joints at Time Points
Description: Forty-four (44) joints were assessed by the Investigator to determine the number of joints that were considered tender or painful. The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be considered for artificial joints). The 44 joints to be assessed were:sternoclavicular, acromioclavicular, shoulder, elbow, wrist (includes radiocarpal, carpal and carpometacarpal considered as one unit), metacarpophalangeals (I, II, III, IV, V), thumb interphalangeal (IP), proximal IPs (II, III, IV, V), knee, ankle, metatarsophalangeals (I, II, III, IV, V).
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Number of joints
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 102 | 105
Number of joints
  Week 2 (N = 100, 102) | -1.99 (0.36) | -1.38 (0.35)
  Week 4 (N = 100, 105) | 1.52 (0.41) | -1.27 (0.39)
  Week 8 (N = 101, 105) | -1.93 (0.41) | -2.02 (0.39)
  Week 12 (N = 101, 105) | -1.55 (0.38) | -1.56 (0.36)
  Week 16 (N = 96, 102) | -1.93 (0.39) | -2.35 (0.49)
  Week 24 (N = 96, 102) | -2.46 (0.43) | -2.83 (0.57)
  Week 32 (N = 96, 102) | -1.96 (0.42) | -3.09 (0.55)
  Week 40 (N = 96, 102) | -2.42 (0.42) | -3.16 (0.53)
  Week 48 (N = 96, 102) | -2.65 (0.42) | -2.95 (0.55)
  Week 56 (N = 96, 102) | -2.44 (0.43) | -3.25 (0.58)
  Week 68 (N = 96, 102) | -2.43 (0.40) | -3.30 (0.61)
  Week 80 (N = 96, 102) | -2.60 (0.43) | -3.07 (0.60)
  Week 92 (N = 96, 102) | -2.45 (0.37) | -3.29 (0.58)
  Week 104 (N = 96, 102) | -2.72 (0.42) | -3.48 (0.58)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0836, ANCOVA; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.32 to 0.08]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.5402, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.02 to 0.54]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.8167, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.69 to 0.87]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.9891, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.72 to 0.73]

47. Secondary Outcome: Mean Change From Baseline in Dactylitis Score at Time Points
Description: Each of the 10 fingers and 10 toes is evaluated for dactylitis. A score of 0, 1, 2 or 3 (where 0 = none, 1= mild, 2 = moderate, 3 = severe) is assigned to each. A total score which can range from 0 to 60 is obtained by adding the scores for the 20 digits
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 108
Units on a scale
  Week 2 (N = 105, 107) | -0.00 (0.03) | 0.02 (0.03)
  Week 4 (N = 105, 108) | -0.09 (0.03) | -0.05 (0.03)
  Week 8 (N = 105, 108) | -0.19 (0.02) | -0.16 (0.02)
  Week 12 (N = 105, 108) | -0.19 (0.08) | -0.21 (0.07)
  Week 16 (N = 100, 104) | -0.21 (0.13) | -0.20 (0.10)
  Week 24 (N = 100, 104) | -0.23 (0.13) | -0.20 (0.10)
  Week 32 (N = 100, 104) | -0.23 (0.13) | -0.21 (0.10)
  Week 40 (N = 100, 104) | -0.22 (0.13) | -0.23 (0.10)
  Week 48 (N = 100, 104) | -0.22 (0.13) | -0.22 (0.09)
  Week 56 (N = 100, 104) | -0.23 (0.13) | -0.22 (0.10)
  Week 68 (N = 100, 104) | -0.20 (0.11) | -0.23 (0.10)
  Week 80 (N = 100, 104) | -0.23 (0.13) | -0.23 (0.10)
  Week 92 (N = 100, 104) | -0.17 (0.10) | -0.23 (0.10)
  Week 104 (N = 100, 104) | -0.23 (0.13) | -0.23 (0.10)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6148, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.08 to 0.05]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2547, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.11 to 0.03]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1208, ANCOVA; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.08 to 0.01]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.8291, ANCOVA; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.13 to 0.17]

48. Secondary Outcome: Changes From Baseline in Maastricht Ankylosing Spondylitis Enthesis Score (MASES) at Time Points
Description: Assessment of enthesitis was performed in the following 7 domains: 1) 1st costochondral joint left and right, 2) 7th costochondral joint left and right, 3) posterior superior iliac spine left and right, 4) anterior superior iliac spine left and right, 5) iliac crest left and right, 6) 5th lumbar spinous process and 7) proximal insertion of Achilles tendon left and right. Each domain was graded for the presence (1) and absence (0) of tenderness yielding total MASES ranging from 0 (no tenderness) to 13 (worst possible score; severe tenderness).
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 105 | 108
Units on a scale
  Week 2 (N = 104, 107) | -0.94 (0.23) | -0.74 (0.22)
  Week 4 (N = 104, 108) | -1.11 (0.27) | -0.65 (0.25)
  Week 8 (N = 104, 108) | -1.39 (0.27) | -1.20 (0.25)
  Week 12 (N = 104, 108) | -1.40 (0.28) | -0.74 (0.26)
  Week 16 (N = 99, 104) | -1.64 (0.24) | -1.50 (0.26)
  Week 24 (N = 99, 104) | -1.78 (0.25) | -1.34 (0.27)
  Week 32 (N = 99, 104) | -1.59 (0.26) | -1.66 (0.28)
  Week 40 (N = 99, 104) | -1.86 (0.26) | -1.62 (0.27)
  Week 48 (N = 99, 104) | -1.79 (0.27) | -1.73 (0.28)
  Week 56 (N = 99, 104) | -2.01 (0.28) | -1.63 (0.30)
  Week 68 (N = 99, 104) | -1.92 (0.27) | -1.73 (0.29)
  Week 80 (N = 99, 104) | -1.99 (0.28) | -1.72 (0.32)
  Week 92 (N = 99, 104) | -2.00 (0.26) | -1.65 (0.30)
  Week 104 (N = 99, 104) | -1.87 (0.28) | -1.77 (0.29)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3536, ANCOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.64 to 0.23]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0769, ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.97 to 0.05]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.4698, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.70 to 0.33]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0167, ANCOVA; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.19 to -0.12]

49. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Concentration Time Points
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 106 | 108
mg/L
  Week 2 (N = 105, 107) | -4.49 (0.71) | -1.46 (0.67)
  Week 4 (N = 105, 108) | -3.61 (1.16) | 0.25 (1.10)
  Week 8 (N = 105, 108) | -4.07 (1.33) | -0.97 (1.27)
  Week 12 (N = 105, 108) | -2.78 (1.14) | 0.65 (1.08)
  Week 16 (N = 100, 104) | -4.84 (1.07) | -3.82 (1.08)
  Week 24 (N = 100, 104) | -4.62 (1.10) | -4.56 (1.04)
  Week 32 (N = 100, 104) | -4.97 (1.01) | -3.88 (1.01)
  Week 40 (N = 100, 104) | -4.88 (1.10) | -4.26 (1.08)
  Week 48 (N = 100, 104) | -4.94 (1.08) | -4.64 (1.06)
  Week 56 (N = 100, 104) | -5.20 (1.04) | -4.59 (1.02)
  Week 68 (N = 100, 104) | -5.03 (1.01) | -3.93 (1.09)
  Week 80 (N = 100, 104) | -4.29 (1.17) | -4.12 (0.99)
  Week 92 (N = 100, 104) | -5.10 (1.06) | -4.44 (1.04)
  Week 104 (N = 100, 104) | -4.28 (1.16) | -3.65 (1.12)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 39, analysis 1]; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.02, 95% CI 2-sided [-4.39 to -1.66]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = -3.86, 95% CI 2-sided [-6.09 to -1.62]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0143, ANCOVA; Mean Difference (Final Values) = -3.04, 95% CI 2-sided [-5.47 to -0.61]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0038, ANCOVA; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-5.23 to -1.02]

50. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Time Points
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hr. A higher rate is consistent with inflammation.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mm/hr
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 101 | 106
mm/hr
  Week 2 (N = 100, 104) | -9.02 (1.61) | -1.30 (1.53)
  Week 4 (N = 100, 106) | -10.00 (1.57) | -3.98 (1.48)
  Week 8 (N = 100, 106) | -10.79 (1.84) | -4.81 (1.76)
  Week 12 (N = 100, 106) | -11.34 (1.80) | -2.68 (1.39)
  Week 16 (N = 95, 102) | -12.75 (2.03) | -9.77 (1.62)
  Week 24 (N = 95, 102) | -14.22 (1.96) | -8.82 (1.77)
  Week 32 (N = 95, 102) | -12.76 (2.04) | -10.13 (1.76)
  Week 40 (N = 95, 102) | -11.49 (2.22) | -10.48 (1.74)
  Week 48 (N = 95, 102) | -12.20 (2.05) | -9.91 (1.90)
  Week 56 (N = 95, 102) | -13.03 (2.18) | -8.91 (1.70)
  Week 68 (N = 95, 102) | -10.80 (2.17) | -9.48 (1.74)
  Week 80 (N = 95, 102) | -10.74 (2.14) | -8.15 (1.74)
  Week 92 (N = 95, 102) | -10.84 (2.28) | -8.79 (1.79)
  Week 104 (N = 95, 102) | -10.51 (2.15) | -5.73 (2.05)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -7.71, 95% CI 2-sided [-10.85 to -4.58]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.12, 95% CI 2-sided [-9.16 to -3.09]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0009, ANCOVA; Mean Difference (Final Values) = -5.78, 95% CI 2-sided [-9.15 to -2.41]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -7.03, 95% CI 2-sided [-10.34 to -3.73]

51. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ)-5D VAS Score Time Points
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: mm
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
mm
  Week 4 (N = 86, 93) | 4.76 (2.20) | 4.77 (2.03)
  Week 8 (N = 85, 93) | 6.66 (2.84) | 3.05 (2.65)
  Week 12 (N = 84, 92) | 9.33 (2.97) | 3.26 (2.77)
  Week 16 (N = 82, 91) | 12.72 (2.16) | 11.56 (2.44)
  Week 24 (N = 82, 90) | 13.21 (2.23) | 16.61 (2.26)
  Week 40 (N = 79, 86) | 16.62 (2.13) | 14.67 (2.64)
  Week 48 (N = 75, 86) | 16.29 (2.37) | 18.72 (2.37)
  Week 68 (N = 72, 82) | 17.26 (2.18) | 17.90 (2.60)
  Week 92 (N = 69, 77) | 16.32 (2.33) | 21.08 (2.73)
  Week 104 (N = 64, 75) | 19.81 (2.45) | 23.69 (2.71)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; With the exception of change from Baseline in the placebo group at Week 12, within group comparisons to baseline for all other treatment groups and time points were <0.001, from paired t-test; Test type: Superiority or Other; p = 0.0370, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4, 8, 12 data only. Week 4; Test type: Superiority or Other; p = 0.9965, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-4.39 to 4.37]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4, 8, 12 data only. Week 8; Test type: Superiority or Other; p = 0.1970, ANCOVA; Mean Difference (Final Values) = 3.61, 95% CI 2-sided [-1.89 to 9.10]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4, 8, 12 data only. Week 12; Test type: Superiority or Other; p = 0.0394, ANCOVA; Mean Difference (Final Values) = 6.07, 95% CI 2-sided [0.30 to 11.84]

52. Secondary Outcome: Change From Baseline in EQ-5D Health State Profile Utility Score at Time Points
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 4 (N = 89, 96) | 0.14 (0.03) | 0.09 (0.03)
  Week 8 (N = 86, 94) | 0.13 (0.04) | 0.08 (0.03)
  Week 12 (N = 85, 93) | 0.19 (0.04) | 0.08 (0.03)
  Week 16 (N = 83, 90) | 0.19 (0.04) | 0.17 (0.03)
  Week 24 (N = 82, 90) | 0.21 (0.03) | 0.20 (0.03)
  Week 40 (N = 79, 86) | 0.24 (0.04) | 0.18 (0.03)
  Week 48 (N= 75, 86) | 0.23 (0.03) | 0.22 (0.03)
  Week 68 (N= 72, 83) | 0.24 (0.04) | 0.22 (0.03)
  Week 92 (N= 69, 78) | 0.24 (0.04) | 0.22 (0.03)
  Week 104 (N= 64, 75) | 0.29 (0.04) | 0.25 (0.03)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.01 at Week 12 and <0.001 thereafter, from paired t-test; Test type: Superiority or Other; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 51, analysis 2]; Test type: Superiority or Other; p = 0.1341, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.02 to 0.21]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 51, analysis 3]; Test type: Superiority or Other; p = 0.0447, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.00 to 0.14]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 51, analysis 4]; Test type: Superiority or Other; p = 0.1345, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.02 to 0.13]

53. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Summary (PCS) at Time Points
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100 = highest level of functioning).
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 4 (N = 89, 96) | 4.04 (0.79) | 2.72 (0.74)
  Week 12 (N = 85, 94) | 6.18 (0.97) | 3.80 (0.91)
  Week 24 (N = 83, 91) | 6.67 (0.93) | 7.29 (0.78)
  Week 48 (N = 77, 86) | 8.03 (0.96) | 8.51 (0.85)
  Week 68 (N = 72, 83) | 8.97 (0.98) | 9.42 (0.94)
  Week 92 (N = 69, 78) | 8.35 (1.15) | 9.28 (0.93)
  Week 104 (N = 65, 75) | 9.98 (1.03) | 10.38 (1.01)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4, 12 data only. Week 4; Test type: Superiority or Other; p = 0.1035, ANCOVA; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-0.27 to 2.90]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 4, 12 data only. Week 12; Test type: Superiority or Other; p = 0.0134, ANCOVA; Mean Difference (Final Values) = 2.38, 95% CI 2-sided [0.50 to 4.26]

54. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary (MCS) at Time Points
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 4 (N = 89, 96) | 2.65 (1.02) | 1.47 (0.94)
  Week 12 (N = 85, 94) | 2.44 (1.29) | 1.58 (1.20)
  Week 24 (N = 83, 91) | 3.52 (1.30) | 4.36 (0.99)
  Week 48 (N = 77, 86) | 3.47 (1.18) | 3.54 (1.07)
  Week 68 (N = 72, 83) | 3.65 (1.23) | 4.44 (1.05)
  Week 92 (N = 69, 78) | 4.18 (1.48) | 4.77 (1.19)
  Week 104 (N= 65, 75) | 4.90 (1.34) | 3.74 (1.06)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.05, from paired t-test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 2]; Test type: Superiority or Other; p = 0.2520, ANCOVA; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [-0.84 to 3.19]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 3]; Test type: Superiority or Other; p = 0.4981, ANCOVA; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [-1.63 to 3.34]

55. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Depression Score at Time Points
Description: This outcome measure is describing the HADS subscale of depression. HADS is a participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms. There is no Total Score for HADS.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 4 (N = 89, 96) | -0.63 (0.33) | -0.39 (0.31)
  Week 12 (N = 85, 94) | -0.45 (0.46) | -0.05 (0.43)
  Week 24 (N = 83, 91) | -1.22 (0.35) | -1.04 (0.31)
  Week 48 (N = 77, 85) | -1.42 (0.38) | -1.04 (0.36)
  Week 68 (N = 72, 82) | -1.61 (0.33) | -1.35 (0.36)
  Week 92 (N = 69, 78) | -1.29 (0.39) | -1.47 (0.38)
  Week 104 (N = 65, 74) | -1.91 (0.40) | -1.61 (0.35)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 2]; Test type: Superiority or Other; p = 0.4621, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.90 to 0.41]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 3]; Test type: Superiority or Other; p = 0.3842, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.28 to 0.50]

56. Secondary Outcome: Change From Baseline in HADS Anxiety Score at Time Points
Description: This outcome measure is describing the HADS subscale of anxiety. HADS is a participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms. There is no Total Score for HADS.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 4 (N = 89, 96) | -0.73 (0.35) | -0.89 (0.32)
  Week 12 (N = 85, 94) | -1.33 (0.45) | -0.81 (0.43)
  Week 24 (N = 83, 91) | -0.89 (0.40) | -1.66 (0.33)
  Week 48 (N = 77, 85) | -1.03 (0.38) | -1.40 (0.34)
  Week 68 (N = 72, 82) | -1.24 (0.39) | -1.76 (0.41)
  Week 92 (N = 69, 78) | -0.96 (0.46) | -2.24 (0.35)
  Week 104 (N = 65, 74) | -1.80 (0.40) | -1.74 (0.39)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 2]; Test type: Superiority or Other; p = 0.6357, ANCOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.52 to 0.86]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 3]; Test type: Superiority or Other; p = 0.2439, ANCOVA; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.39 to 0.36]

57. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score at Time Points
Description: ASQoL is a questionnaire that assesses disease-specific quality of life (QoL). It consists of 18 statements that are relevant to the physical and mental conditions for a participant with Ankylosing Spondylitis (AS): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each statement is answered by the participant as a 'Yes' (scored as 1) or 'No' (scored as 0). All item scores are summed to give a total score. Total score can range from 0 (good QoL) to 18 (poor QoL).
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 96
Units on a scale
  Week 12 (N = 88, 94) | -1.93 (0.54) | -1.42 (0.51)
  Week 24 (N = 83, 91) | -3.12 (0.47) | -3.16 (0.41)
  Week 48 (N = 77, 86) | -3.74 (0.49) | -3.67 (0.43)
  Week 68 (N = 72, 83) | -4.04 (0.48) | -4.10 (0.46)
  Week 92 (N = 69, 77) | -4.00 (0.52) | -4.10 (0.53)
  Week 104 (N = 65, 73) | -4.74 (0.54) | -3.99 (0.54)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Descriptive analysis was carried out for Week 12 data only; Test type: Superiority or Other; p = 0.3286, ANCOVA; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.55 to 0.52]

58. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Work Instability Index (AS-WIS) Score at Time Points
Description: The AS-WIS is a 20 item questionnaire to assess work disability and risk of unemployment due to AS. Higher scores indicate greater work impairment and instability that results from a mismatch between an individual's ability levels given their AS and their job. Each question is assigned a score of 1 for a response of "True" and 0 for a response of "Not True". All item scores are summed to give a total score that can range from 0 to 20. If a subject has ≥ 5 missing responses (ie more than 20%), then a total score is not calculated. For subjects with ≥ 1 but ≤ 4 missing responses, the total score is calculated as follows: T=20x/(20-m) where: T is the total score, x is the total score for the items answered and n is the number of non-missing items.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 87 | 91
Units on a scale
  Week 12 (N = 81, 84) | -2.36 (0.58) | -1.58 (0.55)
  Week 24 (N = 74, 75) | -3.16 (0.58) | -2.71 (0.60)
  Week 48 (N = 66, 75) | -3.61 (0.63) | -4.01 (0.59)
  Week 68 (N = 60, 66) | -4.50 (0.64) | -5.08 (0.71)
  Week 92 (N = 57, 60) | -4.35 (0.76) | -5.27 (0.71)
  Week 104 (N = 55, 62) | -4.78 (0.68) | -5.23 (0.74)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.1829, ANCOVA; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.93 to 0.37]

59. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Percent Work Time Missed Due to Health Problems at Time Points
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated:
  Percent work time missed due to health problem: Q2/(Q2+Q4). The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 62 | 62
Units on a scale
  Week 2 (N = 56, 59) | 2.83 (3.64) | 0.46 (3.58)
  Week 4 (N = 57, 59) | 1.74 (3.35) | 0.12 (3.25)
  Week 8 (N = 53, 53) | 4.19 (4.13) | 0.67 (4.15)
  Week 12 (N = 53, 55) | -0.19 (4.36) | -4.93 (4.25)
  Week 16 (N = 53, 52) | -1.35 (3.34) | -2.03 (4.92)
  Week 24 (N = 47, 47) | -0.71 (3.40) | -7.39 (4.61)
  Week 32 (N = 48, 46) | -4.06 (3.02) | -9.76 (4.12)
  Week 40 (N= 50, 50) | -2.16 (4.15) | -9.23 (3.73)
  Week 48 (N= 48, 47) | -5.04 (2.33) | -6.12 (3.60)
  Week 56 (N= 44, 49) | -3.99 (2.77) | -9.11 (3.79)
  Week 68 (N= 44, 44) | -2.41 (3.19) | -7.51 (3.69)
  Week 80 (N= 43, 44) | 2.92 (2.45) | -9.96 (4.21)
  Week 92 (N= 45, 44) | -1.81 (3.31) | -8.42 (4.29)
  Week 104 (N= 42, 43) | -6.35 (3.45) | -10.44 (4.74)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.05, from paired t-test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5226, ANCOVA; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [-4.95 to 9.68]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.6232, ANCOVA; Mean Difference (Final Values) = 1.62, 95% CI 2-sided [-4.90 to 8.14]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.3877, ANCOVA; Mean Difference (Final Values) = 3.52, 95% CI 2-sided [-4.53 to 11.57]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.2402, ANCOVA; Mean Difference (Final Values) = 4.74, 95% CI 2-sided [-3.22 to 12.69]

60. Secondary Outcome: Change From Baseline in WPAI: Percent Impairment While Working Due to Health Problems at Time Points
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated:
  Percent impairment while working due to health problem: Q5/10. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 59 | 58
Units on a scale
  Week 2 (N = 53, 56) | -11.47 (3.71) | -2.28 (3.67)
  Week 4 (N = 52, 55) | -8.88 (3.66) | -3.81 (3.54)
  Week 8 (N = 47, 50) | -12.74 (3.94) | -6.48 (3.90)
  Week 12 (N = 48, 50) | -21.22 (4.74) | -12.09 (4.70)
  Week 16 (N = 49, 46) | -16.53 (3.69) | -16.09 (2.97)
  Week 24 (N = 46, 43) | -16.52 (4.66) | -18.84 (3.35)
  Week 32 (N = 46, 43) | -18.04 (3.76) | -15.81 (3.45)
  Week 40 (N = 45, 47) | -22.89 (4.04) | -19.36 (2.92)
  Week 48 (N = 45, 47) | -22.22 (3.55) | -16.60 (3.64)
  Week 56 (N = 42, 46) | -23.81 (3.90) | -20.43 (3.33)
  Week 68 (N = 43, 43) | -22.33 (3.96) | -22.09 (3.39)
  Week 80 (N = 42, 41) | -24.29 (4.06) | -21.95 (3.60)
  Week 92 (N = 42, 41) | -23.57 (3.47) | -19.27 (3.07)
  Week 104 (N = 40, 40) | -25.50 (3.69) | -22.50 (3.54)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001 at Week 16 and thereafter, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0193, ANCOVA; Mean Difference (Final Values) = -9.19, 95% CI 2-sided [-16.85 to -1.52]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.1730, ANCOVA; Mean Difference (Final Values) = -5.08, 95% CI 2-sided [-12.41 to 2.26]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1224, ANCOVA; Mean Difference (Final Values) = -6.26, 95% CI 2-sided [-14.23 to 1.71]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0461, ANCOVA; Mean Difference (Final Values) = -9.14, 95% CI 2-sided [-18.11 to -0.16]

61. Secondary Outcome: Changes From Baseline in WPAI - Activity Impairment Due to Health Problems at Time Points
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated:
  Percent activity impairment due to health problem: Q6/10. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 95
Units on a scale
  Week 2 (N = 89, 94) | -10.70 (2.80) | -4.73 (2.61)
  Week 4 (N = 89, 95) | -11.52 (2.45) | -8.42 (2.28)
  Week 8 (N = 86, 93) | -18.35 (3.15) | -11.68 (2.96)
  Week 12 (N = 85, 92) | -18.92 (3.35) | -12.07 (3.14)
  Week 16 (N = 82, 90) | -19.88 (2.77) | -22.33 (2.69)
  Week 24 (N = 82, 89) | -20.61 (3.14) | -23.15 (2.31)
  Week 32 (N = 78, 86) | -20.26 (2.96) | -22.09 (2.58)
  Week 40 (N = 77, 85) | -27.14 (2.85) | -24.00 (2.36)
  Week 48 (N = 74, 85) | -24.46 (2.93) | -22.12 (2.85)
  Week 56 (N = 74, 84) | -25.00 (2.80) | -25.71 (2.44)
  Week 68 (N = 72, 82) | -26.53 (2.95) | -25.73 (2.73)
  Week 80 (N = 69, 77) | -27.39 (3.17) | -27.66 (2.97)
  Week 92 (N = 69, 77) | -26.96 (3.32) | -25.97 (2.81)
  Week 104 (N = 65, 73) | -30.77 (3.01) | -28.36 (2.87)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0372, ANCOVA; Mean Difference (Final Values) = -5.97, 95% CI 2-sided [-11.58 to -0.36]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.2126, ANCOVA; Mean Difference (Final Values) = -3.10, 95% CI 2-sided [-7.98 to 1.79]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.0330, ANCOVA; Mean Difference (Final Values) = -6.66, 95% CI 2-sided [-12.79 to -0.54]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0397, ANCOVA; Mean Difference (Final Values) = -6.85, 95% CI 2-sided [-13.38 to -0.33]

62. Secondary Outcome: Changes From Baseline in WPAI - Overall Work Impairment Due to Health Problems at Time Points
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days. The questions are: Q1 = currently employed. Q2 = hours missed due to health problems. Q3 = hours missed other reasons. Q4 = hours actually worked. Q5 = degree health affected productivity while working (0-10 scale). Q6 = degree health affected regular activities (0-10 scale). Subscale scores are calculated:
  Percent overall work impairment due to health problem:
  Q2/(Q2+Q4)+[(1-Q2/(Q2+Q4))*(Q5/10)]. The computed percentage range for each sub-scale is 0-100, where higher numbers indicate greater impairment and less productivity.
Time Frame: Baseline to Week 104
Population: as for outcome 7
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 58 | 58
Units on a scale
  Week 2 (N = 51, 56) | -7.43 (3.81) | 0.86 (3.74)
  Week 4 (N = 52, 55) | -7.07 (3.72) | -1.82 (3.59)
  Week 8 (N = 47, 49) | -10.32 (4.04) | -4.35 (4.09)
  Week 12 (N = 48, 50) | -20.77 (4.94) | -12.09 (4.89)
  Week 16 (N = 49, 46) | -16.30 (3.83) | -16.39 (2.86)
  Week 24 (N = 45, 43) | -14.85 (4.52) | -18.59 (3.68)
  Week 32 (N = 46, 43) | -17.59 (3.79) | -16.53 (3.33)
  Week 40 (N = 45, 47) | -23.74 (4.15) | -20.52 (3.03)
  Week 48 (N = 45, 45) | -23.03 (3.61) | -17.54 (3.87)
  Week 56 (N = 42, 46) | -23.60 (4.10) | -21.39 (3.43)
  Week 68 (N = 43, 42) | -21.90 (4.26) | -22.27 (3.46)
  Week 80 (N = 42, 41) | -20.66 (4.15) | -23.10 (3.80)
  Week 92 (N = 42, 41) | -24.00 (3.52) | -19.39 (3.24)
  Week 104 (N = 40, 40) | -25.76 (3.73) | -23.01 (3.80)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Within group comparisons to baseline were <0.001 at Week 16 and at Week 32 and thereafter, from paired t test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0382, ANCOVA; Mean Difference (Final Values) = -8.29, 95% CI 2-sided [-16.12 to -0.46]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 4Secondary and supportive analyses were performed at 2-sided alpha = 0.05 significance level. No adjustment for multiple testing was made. Comparative analysis was carried out for Week 2, 4, 8, 12 data only. Week 4; Test type: Superiority or Other; p = 0.1648, ANCOVA; Mean Difference (Final Values) = -5.25, 95% CI 2-sided [-12.69 to 2.19]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1476, ANCOVA; Mean Difference (Final Values) = -5.98, 95% CI 2-sided [-14.11 to 2.15]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority or Other; p = 0.0687, ANCOVA; Mean Difference (Final Values) = -8.68, 95% CI 2-sided [-18.03 to 0.68]

63. Secondary Outcome: Change From Baseline in Multidimensional Fatigue Inventory (MFI) Score at Time Points
Description: The MFI is a 20-item questionnaire that evaluates several aspects of fatigue. The General Fatigue Item is disclosed here. The general fatigue item contains four items, two of which are indicative for fatigue and two items contra-indicative for fatigue. Indicative items (eg, "I tire easily") are formulated in such a way that a high score suggests a high degree of fatigue. In case of contra-indicative items (eg, "I feel fit") a high score indicates a low degree of fatigue. Each item is scored on a 5-point numeric rating scale anchored at each end by "Yes, that is true" (scored 1) to "No, that is not true" (scored 5). Scoring for the MFI is done in such a way that higher scores indicate greater fatigue. Therefore, the items indicative for fatigue need to be recoded (1=5, 2=4, 3=3, 4=2, 5=1). For each scale a total score is calculated by summation of the scores of the individual items. Scores can range from the minimum of 4 to the maximum of 20. MFI-20 scale is copyrighted.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 95
Units on a scale
  Week 4 (N = 89, 95) | -1.08 (0.38) | -0.64 (0.36)
  Week 12 (N = 85, 93) | -1.34 (0.42) | -1.08 (0.39)
  Week 24 (N = 83, 89) | -1.67 (0.37) | -2.69 (0.40)
  Week 48 (N = 77, 85) | -2.01 (0.39) | -2.84 (0.39)
  Week 68 (N = 72, 82) | -1.79 (0.42) | -3.01 (0.45)
  Week 92 (N = 69, 77) | -2.74 (0.40) | -3.18 (0.52)
  Week 104 (N = 65, 73) | -3.26 (0.46) | -3.04 (0.50)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 2]; Test type: Superiority or Other; p = 0.2578, ANCOVA; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-1.21 to 0.33]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 3]; Test type: Superiority or Other; p = 0.4334, ANCOVA; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.21 to 0.52]

64. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale Score From Baseline to Week 104
Description: The MOS sleep scale consists of 12 items to measure 6 sleep dimensions: initiation (time to fall asleep), quantity (hours of sleep each night), maintenance, respiratory problems, perceived adequacy, somnolence (the last 4 items reported using a 6-item Likert scale ranging from 1 [all of the time] to 6 [none of the time]). The raw scores ranging from 1 to 6 are transformed to scores ranging from 0 to 100 before the indices are calculated. Therefore the reported scores, consisting of means of converted items, also range from 0 to 100. However, two indexes can be derived: Sleep problems index I (short form) and sleep problems index II (long form). Additional subscales can be derived: sleep disturbance, snoring, awaken shortness of breath or headache, sleep adequacy, sleep somnolence, sleep quantity, and optimal sleep. However, data for two indexes and additional subscales is not reported.
Time Frame: Baseline to Week 104
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 90 | 95
Units on a scale
  Week 4 (N = 89, 94) | -2.35 (1.59) | -0.85 (1.50)
  Week 12 (N = 85, 93) | -6.01 (2.00) | -4.10 (1.88)
  Week 24 (N = 83, 89) | -11.01 (2.64) | -14.34 (2.28)
  Week 32 (N = 78, 86) | -13.17 (2.30) | -17.06 (2.42)
  Week 48 (N = 76, 85) | -11.97 (2.60) | -17.57 (2.23)
  Week 68 (N = 71, 82) | -10.40 (2.56) | -15.50 (2.49)
  Week 104 (N = 66, 76) | -17.92 (2.78) | -15.61 (2.66)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; All within group comparisons to baseline were <0.001, from paired t-test; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 2]; Test type: Superiority or Other; p = 0.3554, ANCOVA; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-4.70 to 1.70]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 53, analysis 3]; Test type: Superiority or Other; p = 0.3350, ANCOVA; Mean Difference (Final Values) = -1.91, 95% CI 2-sided [-5.82 to 1.99]

65. Secondary Outcome: Percentage of Participants With Minimally Clinically Important Improvement (MCII) at Time Points
Description: The MCII asks participants to rate the level of improvement they have experienced in the 48 hours compared to when they started the study. Response options are "Improved - less pain", "No change", and "Worse - more pain." If the participant indicates that improvement has occurred, then they are asked to indicate how important that improvement is to them from "Not at all important" to "Very important'.
Time Frame: Weeks 12 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 88 | 94
Percentage of participants
  Week 12 (N = 88, 94) | 59.09 | 44.68
  Week 104 (N = 75, 79) | 76.00 | 81.01
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 57, analysis 2]; Test type: Superiority or Other; p = 14.41, ANCOVA; Mean Difference (Final Values) = 14.41, 95% CI 2-sided [0.04 to 28.78]

66. Secondary Outcome: Percentage of Participants Achieving Patient Acceptable Symptom State (PASS) at Time Points
Description: PASS is defined as a symptom state that the participants consider acceptable.
Time Frame: Weeks 12 and 104
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 88 | 94
Percentage of participants
  Week 12 (N = 88, 94) | 72.73 | 61.70
  Week 104 (N = 74, 80) | 79.73 | 88.75
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 57, analysis 2]; Test type: Superiority or Other; p = 0.1285, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 11.03, 95% CI 2-sided [-2.51 to 24.56]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent until Week 104 visit.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Etanercept: Participants were treated with etanercept subcutaneous injection weekly plus stable background NSAID at optimal anti-inflammatory dose for 12 weeks (double-blind period).
- Placebo: Participants were treated with placebo subcutaneous injection weekly plus stable background NSAID at optimal anti-inflammatory dose for 12 weeks (double-blind period).
Arm/Group | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 9/111 | 8/113
Other Adverse Events (participants affected / at risk) | 86/111 | 87/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=111) | Placebo (N=113)
Myocarditis (Cardiac disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Anal abscess (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=111) | Placebo (N=113)
Uveitis (Eye disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 9
Nausea (Gastrointestinal disorders) | 2 | 7
Injection site erythema (General disorders) | 8 | 6
Injection site reaction (General disorders) | 7 | 6
Bronchitis (Infections and infestations) | 7 | 7
Gastroenteritis (Infections and infestations) | 8 | 7
Influenza (Infections and infestations) | 7 | 7
Nasopharyngitis (Infections and infestations) | 26 | 23
Pharyngitis (Infections and infestations) | 5 | 8
Sinusitis (Infections and infestations) | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Headache (Nervous system disorders) | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.